### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | nation Type : Reporting and Analysis Plan (RAP) | |

| Title | : | Reporting and Analysis Plan for Study 204959: An open-label, single arm, repeat dose, multi-centre study to evaluate the use of an autoinjector for the subcutaneous administration of mepolizumab in subjects with severe eosinophilic asthma. |
|---|---|---|
| Compound Number | ŀ | SB-240563 |
| Effective Date | : | 30-NOV-2017 |

## **Description:**

• The purpose of this RAP is to describe the planned analyses and associated data displays to be included in the Clinical Study Report for Protocol 204959.

• This RAP defines the content of the final Statistical Analysis Complete (SAC) deliverable

## **RAP Author(s):**

| Approver | Date | Approval Method |
|----------------------------------------|----------------|-----------------|
| PPD | 16-NOV-2017 | eSignature |
| Statistics Leader, Clinical Statistics | 10-110 V -2017 | CSignature |

Copyright 2017 the GlaxoSmithKline (GSK) group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

## **RAP Team Approvals:**

| Approver | Date | Approval Method |
|----------------------------------------------|-------------|-----------------|
| Director, Clinical Pharmacology | 17-NOV-2017 | eSignature |
| PPD Product Physician Lead | 30-NOV-2017 | email |
| Clinical Investigational Lead | 17-NOV-2017 | eSignature |
| Global Clinical Safety and Pharmacovigilance | 16-NOV-2017 | eSignature |
| Clinical Operations | 21-NOV-2017 | eSignature |
| Data Quality Lead | 16-NOV-2017 | eSignature |
| Programmer/Analyst, Clinical Programming | 22-NOV-2017 | eSignature |
| Medical Writer | 14-NOV-2017 | email |

## **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|--------------------------------|-------------|-----------------|
| Director, Clinical Programming | 14-NOV-2017 | email |
| Director, Clinical Statistics | 16-NOV-2017 | eSignature |

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | DDUCTION | 5 |
| 2. | SUMM<br>2.1.<br>2.2.<br>2.3.<br>2.4. | MARY OF KEY PROTOCOL INFORMATION | 5<br>5<br>7 |
| 3. | PLANI<br>3.1.<br>3.2. | NED ANALYSIS<br>Interim Analyses<br>Final Analyses | 9 |
| 4. | ANAL`<br>4.1. | YSIS POPULATIONSProtocol Deviations | |
| 5. | | Methods for Handling Centres Multiple Comparisons and Multiplicity Handling of Missing Data Data Display Standards 5.4.1. Study Treatment Descriptors 5.4.2. Autoinjector Label Descriptors 5.4.3. Sub-group Display Descriptors Other Considerations for Data Analysis and Data Handling Conventions | 1111121212 |
| 6. | STUD | Y POPULATION ANALYSES | 14 |
| 7. | ANAL`<br>7.1.<br>7.2. | YSES TO EVALUATE AUTOINJECTOR<br>Primary Analysis<br>Secondary Analyses | 15 |
| 8. | PHAR | MACOKINETIC ANALYSES | 17 |
| 9. | BLOO | D EOSINOPHILS | 18 |
| 10. | EXAC | ERBATIONS | 18 |
| 11. | | TY ANALYSES Adverse Event Analyses 11.1.1. Adverse Events of Special Interest Clinical Laboratory Analyses Other Safety Analyses 11.3.1. Injection Pain Assessment | 19<br>19<br>19 |
| 12. | IMMUI<br>12.1. | NOGENICITY ANALYSES Overview of Immunogenicity Analyses | |

### CONFIDENTIAL

| 20 | 1 | 0 | ⊏ | 0 |
|------|----|---|---|---|
| _ ZU | 14 | м | O | 3 |

| 13. | REFE | RENCES | 21 |
|---|---|---|---|
| 14 | APPF | NDICES | 22 |
| | 14.1. | | |
| | | 14.1.1. Protocol Defined Time & Events | |
| | 14.2. | Appendix 2: Study Phases and Treatment Emergent Adverse | |
| | | Events | 27 |
| | | 14.2.1. Treatment Phases | |
| | | 14.2.1.1. Treatment Phases for Adverse Events | |
| | | 14.2.1.2. Treatment Phases for Exacerbations | |
| | 14.3. | | |
| | | 14.3.1. Baseline Definition & Derivations | |
| | | 14.3.1.1. Baseline Definitions | 28 |
| | | 14.3.1.2. Derivations and Handling of Missing Baseline | |
| | | Data | 28 |
| | | 14.3.2. Reporting Process & Standards | |
| | 14.4. | Appendix 4: Derived and Transformed Data | 31 |
| | | 14.4.1. General | 31 |
| | | 14.4.2. Study Population | |
| | | 14.4.3. Evaluation of Autoinjector | |
| | | 14.4.4. Safety | |
| | 14.5. | Appendix 5: Reporting Standards for Missing Data | |
| | | 14.5.1. Premature Withdrawals | |
| | | 14.5.2. Handling of Missing Data | |
| | | 14.5.3. Handling of Missing Dates | 34 |
| | | 14.5.4. Handling of Missing Time Point for Assessment of | |
| | | Injection Pain | 34 |
| | 14.6. | Appendix 6: Values of Potential Clinical Importance | 35 |
| | | 14.6.1. Laboratory Values of Potential Clinical Concern | |
| | 14.7. | Appendix 7: Abbreviations & Trade Marks | |
| | | 14.7.1. Abbreviations | |
| | 440 | 14.7.2. Trademarks | |
| | 14.8. | Appendix 8: List of Data Displays | |
| | | 14.8.1. Study Population Tables | |
| | | 14.8.3. Pharmacokinetic Analyses | |
| | | 14.8.4. Pharmacodynamic Analyses | |
| | | 14.8.5. Exacerbations | |
| | | 14.8.7. Immunogenicity | |
| | | 14.8.8. ICH and Other Listings | |
| | 1 <u>/</u> 0 | Appendix 9: Example Mock Shells for Data Displays | |
| | 1 <del>7</del> .J. | Appendia 3. Lagripie ivider diferis IUI Dala Displays | <del>U</del> J |

### 1. INTRODUCTION

The purpose of this RAP is to describe the analyses to be included in the Clinical Study Report (CSR) for Protocol 204959:

| Protocol Revision C | Protocol Revision Chronology: | |
|---|---|---|
| 2016N275054_01 | 18-AUG-2016 | Original |
| 2016N275054_03 | 13-OCT-2016 | Amendment No. 1: Updated to refine the criteria for a successful injection, and amend exclusion criteria 7 and 15. |
| 2016N275054_04 | 15-FEB-2017 | Amendment No. 2: Updated to include a change to the labelling of the autoinjector in some geographical regions, and amend inclusion criteria 5. |

All subjects in this study were recruited after the effective date of Protocol Amendment 2.

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

An additional analysis population was defined for reporting screen failures and inclusion exclusion criteria deviations. This population is described in Section 4.

There are no other changes to the protocol defined statistical analysis plan.

## 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoint |
| To assess the use of the combination product, mepolizumab liquid drug product in autoinjector, for the subcutaneous self-administration of mepolizumab by subjects with severe eosinophilic asthma. | Proportion of subjects successfully able to self-<br>administer their observed third dose at Week 8. |
| Secondary Objectives | Secondary Endpoints |
| To assess the use of mepolizumab<br>liquid drug product in autoinjector<br>outside the clinic setting. | Proportion of subjects successfully able to<br>self-administer their unobserved second dose<br>outside the clinic setting at Week 4 |
| Other Objectives | Other Endpoints |
| To assess the use of mepolizumab<br>liquid drug product in autoinjector<br>both inside and outside of the clinic<br>setting. | <ul> <li>Proportion of subjects successfully able to<br/>self-administer their observed first dose at Week 0</li> <li>Proportion of subjects successfully able to<br/>self-administer both their unobserved second dose</li> </ul> |

| Objectives | Endpoints |
|---|---|
| | <ul> <li>and observed third observed dose at Weeks 4 and 8</li> <li>Proportion of subjects successfully able to self-administer all three doses at Weeks 0, 4 and 8</li> </ul> |
| To evaluate autoinjector use & functionality. | Device usability/functionality questionnaire completed at the End of Study/Early Withdrawal Visit |
| To evaluate any autoinjector injection errors/failures related to use or device performance. | <ul> <li>Investigator evaluation of user/device errors</li> <li>Root cause analysis of each unsuccessful injection</li> </ul> |
| To characterise the subject<br>experience of using the<br>mepolizumab liquid drug product in<br>autoinjector. | Subject Exit Interviews completed over the telephone after the End of Study/Early Withdrawal Visit |
| To assess mepolizumab plasma<br>trough concentrations (C <sub>trough</sub> )<br>following the SC administration of<br>mepolizumab liquid drug product in<br>autoinjector. | Mepolizumab plasma trough concentrations (C <sub>trough</sub> ) at Weeks 4, 8 and 12 |
| To assess the pharmacodynamic<br>(PD) effect following the SC<br>administration of mepolizumab<br>liquid drug product in autoinjector. | Ratio to baseline of blood eosinophils at Weeks 4, 8 and 12 |
| To assess the frequency of asthma exacerbations. | Incidence of asthma exacerbations, expressed as<br>the number of subjects with at least one<br>exacerbation |
| Safety Objectives | Safety Endpoints |
| To evaluate the safety and tolerability of mepolizumab liquid drug product in autoinjector. | Incidence and frequency of Adverse Events (AEs) / Serious Adverse Events (SAEs) including systemic reactions and local injection site reactions |
| | Clinically significant change in haematological and/or clinical chemistry parameters |
| | Vital signs |
| | 12-lead electrocardiogram (ECG) |
| | Incidence of immunogenicity |
| | Level of self-reported pain immediately following,1-<br>and 24-hours following each injection (patient diary) |

## 2.3. Study Design



| Overview of Study Desi | Overview of Study Design and Key Features |
|---|---|
| | or |
| | Subjects not receiving mepolizumab treatment at Visit 1 meeting additional criteria of asthma of eosinophilic phenotype requiring regular treatment with high dose inhaled corticosteroids (ICS)¹ in the 12 months prior to Visit 1, current treatment with an additional controller medication besides ICS for at least 3 months, and with one or more exacerbations in the 12 months prior to Visit 1. Subjects are permitted to be enrolled without continuous high dose ICS, following discussion with the GSK Medical Monitor, providing the subject was receiving continuous ICS and the Investigator attests that the subject should have been treated with high dose ICS but this was precluded by financial or tolerance issues. |
| Dosing | 100 mg mepolizumab SC every 4 weeks (3 administrations) in thigh, abdomen or upper arm (caregiver only). |
| Treatment<br>Assignment | <ul> <li>All subjects will receive the same treatment.</li> <li>Autoinjector labelling will differ dependent on the country: subjects in the US, UK and Australia will use an autoinjector with a pictogram plus standard labelling elements, subjects in all other countries will use an autoinjector with standard labelling elements only.</li> </ul> |
| Interim Analysis | No interim analysis is planned. |
| Time and events | See Appendix 1: Time & Events. |

## 2.4. Statistical Hypotheses

The study is designed to descriptively evaluate the successful use of the mepolizumab liquid drug product in autoinjector for self-administration by subjects with severe eosinophilic asthma.

No formal statistical hypothesis testing is planned. Separate summaries of successful use will be provided for the group of subjects using labelling that includes a pictogram plus standard labelling elements, and the group of subjects using the standard labelling without the pictogram. The number and percentage of subjects successfully able to self-administer each mepolizumab dose will be reported, including 95% confidence intervals (CI). No comparison between the labels will be performed.

## 3. PLANNED ANALYSIS

## 3.1. Interim Analyses

No interim analysis is planned.

## 3.2. Final Analyses

The final planned analyses will be performed after the completion of the following steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze (DBF) has been declared by Data Management.

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects<br>Enrolled (ASE) | All subjects for whom a record exists in the data base. | Pre-screen and screen failures |
| All Subjects<br>(Safety) | All enrolled subjects attempting at least one self-administration of mepolizumab. | <ul> <li>Endpoints relating to<br/>autoinjector use and<br/>functionality,<br/>including primary<br/>endpoint</li> <li>Study Population</li> <li>Safety</li> </ul> |
| Pharmacokinetic<br>(PK) | All enrolled subjects attempting at least one self-administration of mepolizumab for whom a PK sample was obtained and analysed. | • PK |
| Pharmacodynamic (PD) | All enrolled subjects attempting at least one self-administration of mepolizumab who had a baseline PD measurement and at least one post-treatment PD measurement. | • PD |

#### NOTES:

• Please refer to Appendix 8: List of Data Displays which details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan (PDMP).
  - o Data will be reviewed prior to DBF to ensure all important deviations are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, subject management or subject assessment) will be summarised and listed.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the electronic case report form (eCRF).

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Methods for Handling Centres

In this multi-centre global study, enrolment will be presented by investigative site within country.

Each autoinjector will have labelling that includes a pictogram plus standard labelling elements, or a standard labelling without the pictogram. Centres in the US, UK and Australia will use labelling that includes a pictogram plus standard labelling elements, while centres in Canada, Germany, Netherlands, Russia and Sweden will use standard labelling without the pictogram. Separate summaries of successful use will be provided for the group of subjects using labelling that includes a pictogram plus standard labelling elements, and the group of subjects using the standard labelling without the pictogram.

## 5.2. Multiple Comparisons and Multiplicity

No formal hypothesis will be tested in the study. Each endpoint will be considered separately and no adjustment for multiplicity will be made.

## 5.3. Handling of Missing Data

In general, analysis will be performed on all available data and no imputation will be performed for missing data. However, if there are withdrawals from study treatment due to issues pertaining to the use of the autoinjector, sensitivity analysis of the primary endpoint will be performed. Missing injection success assessments for subjects withdrawing from study treatment due to issues with the autoinjector will be included in the analysis as injection success assessments classed as "not attempted" on the eCRF for subjects withdrawing from study treatment due to issues with the autoinjector will also be included in this analysis as injection failures.

## 5.4. Data Display Standards

## 5.4.1. Study Treatment Descriptors

| RandAll NG | Data Displays for Reporting | |
|----------------|-----------------------------|-------|
| Description | Description | Order |
| Not applicable | Liquid Autoinjector | 1 |

## 5.4.2. Autoinjector Label Descriptors

Analyses to evaluate the autoinjector will be reported separately for the group of subjects using autoinjectors with labelling that includes a pictogram plus standard labelling elements, and the group of subjects using the standard labelling without the pictogram. Listings of autoinjector evaluation data will include the following label descriptions:

| | Reporting Group Descriptions – Autoinjector Label | | | |
|---|---|---|---|---|
| RandAll NG | | Country | Data Displays for Reporting | |
| Code | Description | Country | Description | Order |
| | | Australia, UK, US | Standard Label + Pictogram | 1 |
| Not applicable | | Canada, Germany,<br>Netherlands,<br>Russia, Sweden | Standard Label | 2 |

## 5.4.3. Sub-group Display Descriptors

| Data Displays for Reporting | | |
|------------------------------------|-----------|---|
| Subgroup Descriptor Category Order | | |
| Baseline Mepolizumab Use | No | 1 |
| | Yes | 2 |
| Injection Site | Abdomen | 1 |
| | Upper Arm | 2 |
| | Thigh | 3 |

# 5.5. Other Considerations for Data Analysis and Data Handling Conventions

Table 1 provides an overview of the appendices within the RAP for outlining other general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| Section 14.1 | Appendix 1: Schedule of Activities |
| | Protocol Defined Time & Events |
| Section 14.2 | Appendix 2: Study Phases and Treatment Emergent Adverse Events |
| | Treatment Phases for Adverse Events |
| | Treatment Phases for Exacerbations |
| Section 14.3 | Appendix 3: Data Display Standards & Handling Conventions |
| | Baseline Definition & Derivations |
| | Reporting Process & Standards |
| Section 14.4 | Appendix 4: Derived and Transformed Data |
| | General |
| | Study Population |
| | Evaluation of Autoinjector |
| | Safety |
| Section 14.5 | Appendix 5: Reporting Standards for Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| | Handling of Missing and Partial Dates |
| Section 14.6 | Appendix 6: Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES

The study population analyses will be based on the "All Subjects (Safety)" population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, concomitant medications and exposure will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 8: List of Data Displays.

#### 7. ANALYSES TO EVALUATE AUTOINJECTOR

- All analyses will be based on the "All Subjects (Safety)" population.
- All analyses to evaluate the autoinjector will be reported separately for the group of subjects using autoinjectors with labelling that includes a pictogram plus standard labelling elements, and the group of subjects using the standard labelling without the pictogram. No comparison between the labels will be performed.

## 7.1. Primary Analysis

The primary endpoint is the proportion of subjects successfully able to self-administer their observed third dose at Week 8.

- The number and percentage of subjects successfully able to self-administer their observed third dose at Week 8 will be summarized together with 95% CI.
- The denominator for the percentage calculation will be the number of subjects attempting an injection at Week 8.
- CI for the percentages will be generated using the Exact (Clopper-Pearson) method for binomial proportions.
- No formal statistical analysis will be conducted and no comparison between labels will be performed.
- If a subject has more than one attempt to self-administer study treatment at Week 8, the first attempt will be included in the primary analysis. The best attempt will also be summarised as a supportive analysis. A separate listing of injection success for subjects who had more than one attempt to self-administer mepolizumab will be provided.
- If there are withdrawals from study treatment due to issues pertaining to the use of the autoinjector, a sensitivity analysis of the primary endpoint will be performed. Missing injection success assessments for subjects withdrawing from study treatment due to issues with the autoinjector will be included in the analysis as injection failures i.e. as unsuccessful attempts to self-administer mepolizumab. Injection success assessments classed as "not attempted" on the eCRF for subjects withdrawing from study treatment due to issues with the autoinjector will also be included in this analysis as injection failures.

Full details of data displays being presented in Appendix 8: List of Data Displays.

## 7.2. Secondary Analyses

The following endpoints will be summarised in the same way as the primary endpoint (Section 7.1).

- The number and percentage of subjects successfully able to self-administer their unobserved second dose at Week 4. The denominator for the percentage calculation will be the number of subjects attempting an injection at Week 4.
- The number and percentage of subjects successfully able to self-administer their observed first dose at Week 0. The denominator for the percentage calculation will be the number of subjects attempting an injection at Week 0.
- The number and percentage of subjects successfully able to self-administer both their unobserved second dose at Week 4 and their observed third dose at Week 8. The denominator for the percentage calculation will be the number of subjects attempting an injection at both Week 4 and Week 8.
- The number and percentage of subjects successfully able to self-administer all three doses at Week 0, 4 and 8. The denominator for the percentage calculation will be the number of subjects attempting all three doses at Week 0, 4 and 8.

Data collected on the observer checklist for in-clinic injections and subject completed checklists for home injections will be summarised. The investigator assessment of user/device errors will be summarised by visit. Device usability/functionality assessed by the subject at the end of the study will also be summarised.

Full details of data displays being presented in Appendix 8: List of Data Displays.

### 8. PHARMACOKINETIC ANALYSES

- The PK analyses will be based on the "PK" population.
- Linear and semi-logarithmic individual mepolizumab plasma concentration-time profiles will be produced for each subject. Time will be relative to the first dose of study treatment. Individual mepolizumab plasma concentration-time profile plots grouped by baseline mepolizumab use and by baseline mepolizumab use and injection site (performed only for the subset of subjects using the same injection site throughout the study) will also be produced.
- Mepolizumab plasma concentrations will be listed and summarised by nominal time and by nominal time and baseline mepolizumab use. Mean (±SD) and median profiles by nominal time and baseline mepolizumab use will be plotted.
- Summaries of mepolizumab plasma concentration-time data will also be produced by baseline mepolizumab use and injection site, and mean (±SD) and median concentration-time profiles by baseline mepolizumab use and injection site will be plotted. These summaries will be performed only for the subset of subjects using the same injection site throughout the study.
- Refer to Appendix 3: Data Handling Conventions, Section 14.3.2 Reporting Process & Standards.

Full details of the data displays to be presented are given in Appendix 8: List of Data Displays.

### 9. BLOOD EOSINOPHILS

- Blood eosinophil analyses will be based on the "Pharmacodynamic" population.
- Blood eosinophil values will be log<sub>e</sub>-transformed prior to summarising. Non-detectable values of 0 GI/L, will be replaced by half of the lowest observed detectable (non-zero) value in the study data set, prior to log transformation.
- Blood eosinophil values will be summarised by visit, and by visit and baseline mepolizumab use.
- Blood eosinophil values will also be summarised by visit, baseline mepolizumab use and injection site. These summaries will be performed only for the subset of subjects using the same injection site throughout the study.
- Absolute and ratio to baseline blood eosinophils will be listed.

Full details of data displays to be presented are given in Appendix 8: List of Data Displays.

## 10. EXACERBATIONS

Analyses of exacerbations will be based on the "All Subjects (Safety)" population. The number and percentage of subjects with at least one on-treatment exacerbation will be summarised. On-treatment exacerbations are defined in Section 14.2.1.2. All exacerbation data will be listed.

#### 11. SAFETY ANALYSES

Analysis of safety data will be based on the 'All Subjects (Safety)" population.

## 11.1. Adverse Event Analyses

Adverse event analyses including the analysis of AEs, SAEs and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 8: List of Data Displays.

### 11.1.1. Adverse Events of Special Interest

Adverse events of special interest (AESIs) are AEs associated with the identified and potential risks of mepolizumab. AESIs reported by the investigator as anaphylaxis reactions, systemic reactions (further categorised by the investigator as either allergic [type I hypersensitivity] or other systemic reactions) and local injection site reactions are collected via targeted eCRF within the study.

AESIs of opportunistic infections, malignancies, serious cardiac, vascular and thromboembolic (CVT) events and serious ischemic events will be identified from a list of relevant preferred terms maintained within a project level reference dataset created based on the MedDRA dictionary available at the time of DBF for this study. Further details of how relevant preferred terms are identified are given in the Program Safety Analysis Plan (PSAP).

Separate summary tables showing the number and percent of subjects with each type of AESI, broken down by preferred term will be created.

For each type of AESI a profile summary table will be produced containing information including, but not limited to, the number of occurrences of the event, event characteristics, time to onset, intensity, outcome and action taken.

Separate listings of AESIs identified by the investigator as anaphylaxis, allergic (type I hypersensitivity), other systemic reactions and local injection site reactions will be produced, as well as listings of opportunistic infections, malignancies, serious CVT events and serious ischemic events.

# 11.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Haematology laboratory tests and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 8: List of Data Displays.

A scatter plot of maximum ALT vs baseline ALT, and maximum ALT vs total bilirubin will be produced. In addition, if any liver stopping or liver monitoring events occur during the study, summaries of liver monitoring/stopping event reporting and hepatobiliary laboratory abnormalities will be produced.

## 11.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 8: List of Data Displays.

### 11.3.1. Injection Pain Assessment

Injection pain assessed immediately after the injection and at 1 and 24 hours post-injection, will be summarised by visit and time point. Summary statistics of the Visual Analogue Scale (VAS) score for injection pain will be presented. Categorical summaries of pain description (sharp/stinging, dull/aching, burning, other), pain relative to expectation (greater than expected, less than expected, as expected) and acceptability of pain will also be summarised. All injection pain data will be listed.

#### 12. IMMUNOGENICITY ANALYSES

## 12.1. Overview of Immunogenicity Analyses

For the immunogenicity assessment, two types of anti-drug antibody (ADA) assays will be performed, a binding antibody assay and a neutralising antibody assay.

For the binding assay, there will be a three tiered analysis: screening, confirmation and titration. The screening assay produces a result of positive or negative relative to a screening cut point. Positive samples continue with the confirmation assay, which also produces a result of positive or negative relative to a confirmation cut point. For positive confirmation samples, a titre value will also be obtained to quantify the degree of binding in a titration assay and the sample will be tested with the neutralising assay, which also reports results as positive or negative.

The binding ADA results at Week 0 and Week 12/Early withdrawal will be summarised by visit. Summary statistics for the titre result at Week 12/Early Withdrawal will also be presented. Summaries will also be produced by visit and baseline mepolizumab use.

A summary of adverse events by Week 12/Early Withdrawal binding ADA result will be produced.

A summary of liquid treatment emergent positive confirmatory binding ADA assays in the subset of subjects who did not have a positive confirmatory binding ADA assay prior to the first dose of liquid study treatment at Week 0 will also be presented.

Neutralising antibody assay results will be summarised by visit, and by visit and baseline mepolizumab use.

Immunogenicity data will be listed for subjects with at least one positive screening binding assay.

## 13. REFERENCES

GlaxoSmithKline Document Number 2016N275054\_04 Study ID 204959. An open-label, single arm, repeat dose, multi-centre study to evaluate the use of an autoinjector for the subcutaneous administration of mepolizumab in subjects with severe eosinophilic asthma (Study 204959). Report Date 15-FEB-2017.

## 14. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 : General Considerations for Data Analyses & Data Handling Conventions | |
| Section 14.1 | Appendix 1: Schedule of Activities |
| | Protocol Defined Time & Events |
| Section 14.2 | Appendix 2: Study Phases and Treatment Emergent Adverse Events |
| | Treatment Phases for Adverse Events |
| | Treatment Phases for Exacerbations |
| Section 14.3 | Appendix 3: Data Handling Conventions |
| | Baseline Definition & Derivations |
| | Reporting Process & Standards |
| Section 14.4 | Appendix 4: Derived and Transformed Data |
| | General |
| | Study Population |
| | Evaluation of Autoinjector |
| | Safety |
| Section 14.5 | Appendix 5: Reporting Standards for Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| | Handling of Missing Dates |
| Section 14.6 | Appendix 6: Values of Potential Clinical Importance |
| Other RAP Ap | Other RAP Appendices |
| Section 14.7 | Appendix 7: Abbreviations & Trade Marks |
| Section 14.8 | Appendix 8: List of Data Displays |
| Section 14.9 | Appendix 9: Example Mock Shells for Data Displays |

# 14.1. Appendix 1: Schedule of Activities

## 14.1.1. Protocol Defined Time & Events

| | Pre-screening Week -6<br>to Week -5a | Screening Week -4<br>to Week -1 | Week 0<br>(Day 1) | Week 4<br>(±7 days) | Week 8<br>(±7 days) | End of Study/ Early Withdrawal <sup>b</sup><br>Week 12 (±7 days) |
|---|---|---|---|---|---|---|
| Visit number | V0 | V1 | V2 | V3 | V4 | V5 |
| Informed consent | X | | | | | |
| Demography/child bearing status assessment | X | | | | | |
| Medical history | | X | | | | |
| Asthma and Exacerbation history | Х | | | | | |
| Asthma Therapy history | Х | | | | | |
| Smoking history | | Х | | | | |
| Parasitic screening <sup>c</sup> | | Х | | | | |
| Prior needle use / self-administration assessment | | Х | | | | |
| Inclusion/Exclusion criteria | | Х | | | | |
| Training session | | | Χd | | | |
| Autoinjector self-administration in clinic | | | Χ | | Χ | |
| Autoinjector self-administration outside of clinic | | | | Xe, f | | |
| Laboratory: | | | | | | |
| Urine pregnancy test | | Х | Χd | Xq | Χq | X |
| Haematology (including eosinophils) <sup>9</sup> / Clinical Chemistry | | Х | Xq | Xq | Xq | Xq |
| Urinalysis | | Х | | | | |
| Immunogenicity | | | Χd | | | Xq |
| PK | | | Χď | Xq | Χq | Xq |
| Pharmacogenetics <sup>h</sup> | | | Χ | | | |
| Physical/Clinical: | | | | | | |
| Vital signs <sup>i</sup> | | Х | Χd | Xq | Χq | X |
| 12-lead ECG | | X | | | | X |
| Physical examination | | X | | | | X |
| Weight | | X | | | | |

| | Pre-screening Week -6<br>to Week -5 <sup>a</sup> | Screening Week -4<br>to Week -1 | Week 0<br>(Day 1) | Week 4<br>(±7 days) | Week 8<br>(±7 days) | End of Study/ Early Withdrawalb<br>Week 12 (±7 days) |
|---|---|---|---|---|---|---|
| Visit number | V0 | V1 | V2 | V3 | V4 | V5 |
| Concomitant Medication | Х | Х | Х | Х | Х | X |
| Asthma Exacerbations | | X | Χ | X | Χ | X |
| Serious Adverse Events <sup>j,k,l</sup> | Χ | X | Χ | Χ | Χ | X |
| Adverse Events <sup>j,k,l</sup> | | | Χ | X | X | X |
| Dispense patient diary | | | Χm | Х | Х | |
| Return/review patient diary | | | | Х | Χ | Xn |
| Dispense autoinjector for self-administration outside of clinic | | | | Х | | |
| Return/ inspect autoinjector following self-<br>administration outside of clinic | | | | | Х | Xn,o |
| Subject completed pain assessment diary (0, 1-and 24hours post dose) | | | Χ | Xf | Х | |
| Autoinjector observer assessment checklist | | | Χ | | X | |
| Subject/caregiver completed autoinjector checklist | | | | Χf | | |
| Assessment of injection success | | | Х | | Хр | |
| Device usability/functionality questionnaire | | | | | | X |
| Exit Interview <sup>q</sup> | | | | | | (X) |

- a. Pre-screening Visit (V0) can occur on the same day as the Screening Visit (V1) but must be completed prior to initiating any Visit 1 procedures; The Pre-screening Visit can be conducted up to a maximum of 2 weeks prior to the Screening Visit.
- b. The Early Withdrawal Visit will occur 4 weeks (±7 days) after last dose of mepolizumab for any subject who withdraws prior to Week 12
- c. Parasitic screening is only required in countries with high-risk or for subjects who have visited high-risk countries in the past 6 months. Sites should use local laboratories.
- d. Perform prior to mepolizumab administration during the study and prior to restarting pre-study mepolizumab treatment on study completion/early withdrawal.
- e. Subjects will be instructed to contact clinical study staff at any time if they have concerns or questions regarding self-administration. They will have the option of returning to the clinical site for further training or assistance with self-administration. Requirement for additional training or assistance will be documented.
- f. Self-administration of mepolizumab using the autoinjector should occur within 24 hours following the clinic visit.
- g. Includes measurement of eosinophil levels for pharmacodynamic analysis at Visits 2, 3, 4 and 5 (Week 0, 4, 8 and 12)
- h. Pharmacogenetic sample may be drawn any time after the respective informed consent form is signed and the subject is enrolled.
- i. Vital signs include temperature, sitting blood pressure, respiratory rate and pulse.

#### CONFIDENTIAL

204959

- j. Any SAEs assessed as related to study participation (e.g., study treatment, protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK concomitant medication, will be recorded from the time a subject consents to participate in the study up to and including any follow up contact. All other AEs/SAEs are recorded from the start of study treatment until the End of Study / Early Withdrawal visit.
- k. Injection site reactions (e.g., induration, erythema, edema, rash, pruritus, pain) are to be recorded on both AE and SAE CRF forms.
- I. Information on systemic reactions and events that meet the anaphylaxis criteria is collected on both AE and SAE CRF forms.
- m. Patient diary should be dispensed prior to administration of injection
- n. For any subject who withdraws prior to Week 12 (V5), patient diary and study drug for self-administration outside of clinic will be returned at the Early Withdrawal visit (if applicable).
- o. Assessment to be completed at the Early Withdrawal visit only if the dose of mepolizumab immediately prior to withdrawal was administered outside of the clinic.
- p. Includes both the injection outside the clinic from Week 4 (V3) and the injection in clinic at Week 8 (V4)
- q. In a subset of subjects only. Completed over the telephone after the End of Study/Early Withdrawal Visit

# 14.2. Appendix 2: Study Phases and Treatment Emergent Adverse Events

## 14.2.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to the first dose of study treatment.

#### 14.2.1.1. Treatment Phases for Adverse Events

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE start date < First dose of study treatment <sup>1</sup> |
| On-Treatment | <ul> <li>First dose of study treatment¹ ≤ AE start date ≤ Last dose of study treatment + 28 days</li> <li>Any AE with missing start date will be assumed to be "On-Treatment".</li> <li>Any AE with partial start date will be assumed to be "On-Treatment" unless there is evidence to the contrary (e.g. month/year of onset is present and is earlier than the month/year of the first dose of study treatment).</li> </ul> |
| Post-Treatment | AE start date > Last dose of study treatment + 28 days |

<sup>1</sup>Note: the first dose of study treatment will be defined as the earliest dosing date/time entered into the eCRF, regardless of whether self-administration of the injection was successful i.e. full dose administered for this dosing occasion.

#### 14.2.1.2. Treatment Phases for Exacerbations

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Exacerbation onset date < First dose of study treatment <sup>1</sup> |
| On-Treatment | • First dose of study treatment¹ ≤ exacerbation onset date ≤ Last dose of study treatment + 28 days |
| | Any exacerbation with missing onset date will be assumed to be "On-Treatment". |
| | Any exacerbation with partial onset date will be assumed to be "On-Treatment" unless there is evidence to the contrary (e.g. month/year of onset is present and is earlier than the month/year of the first dose of study treatment). |
| Post-Treatment | Exacerbation onset date > Last dose of study treatment + 28 days |

<sup>1</sup>Note: the first dose of study treatment will be defined as the earliest dosing date/time entered into the eCRF, regardless of whether self-administration of the injection was successful i.e. full dose administered for this dosing occasion.

## 14.3. Appendix 3: Data Handling Conventions

#### 14.3.1. Baseline Definition & Derivations

#### 14.3.1.1. Baseline Definitions

- Baseline will be defined for all subjects in the 'All Subjects (Safety)' population.
- The baseline values for each assessment will be the latest available assessment prior to administration of mepolizumab at Visit 2.

## 14.3.1.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |
| Ratio to Baseline | = Visit Value / Baseline |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 14.3.1.1 will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.

#### 14.3.2. Reporting Process & Standards

| Reporting Process | |
|---|---|
| Software | |
| The currently s | The currently supported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Area : sb240563/mid204959 | |
| Analysis Datasets | |

- Analysis Data Model (ADaM) datasets will be created according to Clinical Data Interchange Standards Consortium (CDISC) standards.
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from System Independent (SI) to Study Data Tabulation Model (SDTM).

#### **Generation of RTF Files**

Rich text format (RTF) files will be generated for the final reporting effort.

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables

#### **Reporting Standards**

- 7.01 to 7.13: Principles Related to Graphics
- Safety and study population displays will be based on the core IDSL templates for these data types.

### **Formats**

• The reported precision (decimal places [DPs]) will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DPs.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings.

#### **Unscheduled Visits**

- Data recorded at an unscheduled visit will be re-assigned in the ADaM data sets to the closest nominal visit at which collection of data was scheduled, unless information already exists at that visit. Unscheduled data re-assigned to a scheduled visit will be reported in summary tables and figures. Unscheduled data that is not re-assigned to a scheduled visit will not be included in summary tables or figures by scheduled visit, with the exception of any unscheduled assessments of injection success which may be included in the summary of "best attempt" investigator assessment of self-administration of study treatment if appropriate see Section 7.1. Unscheduled data that is not re-assigned to a scheduled visit will be considered in the derivation of baseline or highest/worst case post-baseline result for the summary tables.
- Data from all unscheduled visits will be included in listings and individual subject figures.

#### **Early Withdrawal Visits**

- Data recorded at the early withdrawal visit will be re-assigned in the ADaM data sets to the
  next scheduled visit, unless information already exists at that visit. Early withdrawal data reassigned to a scheduled visit will be reported at that visit in summary tables and figures. Early
  withdrawal visit data that is not re-assigned to a scheduled visit will not be included in summary
  tables or figures by scheduled visit. However early withdrawal data that is not re-assigned to a
  scheduled visit will be considered in the derivation of highest/worst case post-baseline result
  for the summary tables.
- Data from all early withdrawal visits will be included in listings and individual subject figures.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharmacokinetic Concentration Data | |
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |

### CONFIDENTIAL

| Reporting Standards | |
|---|---|
| Summary Statistics | Summary Statistics Assign zero to non-quantifiable (NQ) values (Refer to GUI_51487 for further details) |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

## 14.4. Appendix 4: Derived and Transformed Data

#### 14.4.1. General

### **Multiple Measurements at One Time Point**

- May arise when unscheduled visits are re-assigned to a nominal visit (see Section 14.3.2). If
  there is data at the nominal visit, the nominal visit data will be used in the summary tables and
  figures, with the exception of any unscheduled assessments of injection success which may be
  included in the summary of "best attempt" investigator assessment of self-administration of
  study treatment if appropriate see Section 7.1. All assessments will be listed.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance (PCI) summary tables.

## **Study Day**

- Calculated as the number of days from the earliest dosing date/time entered into the eCRF, regardless of whether self-administration of the injection was successful i.e. full dose administered for this dosing occasion.
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Visit 2 Date → Study Day = Ref Date Visit 2 Date</li>
  - Ref Data ≥ Visit 2 Date → Study Day = Ref Date (Visit 2 Date) + 1

## 14.4.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth day and month will be imputed '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Age will be calculated relative to the date of the screening visit (Visit 1).

#### **Body Mass Index (BMI)**

• Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

#### **Disease Duration**

Calculated in years as Number of Years + (Number of Months)/12

#### **Extent of Exposure**

 Number of months of exposure to liquid mepolizumab during this study will be calculated based on the formula:

# Duration of Exposure (Months) = (Date of Last Dose of Study Treatment – Date of First Dose of Study Treatment + 29) × 12/365.25

 The first dose of study treatment will be defined as the earliest dosing date/time entered into the eCRF, regardless of whether self-administration of the injection was successful i.e. full dose administered for this dosing occasion.

## 14.4.3. Evaluation of Autoinjector

#### Time from removal of autoinjector from storage to injection

Calculated in minutes as Time of Injection – Time Autoinjector Removed from Storage

## 14.4.4. Safety

#### **Adverse Events**

#### **Drug Related AEs**

AEs with relationship marked 'YES' or relationship missing.

### AEs Leading to Permanent Discontinuation from Study Treatment or Withdrawal from the Study

AEs with action marked "Study treatment withdrawn" or withdrawn from study status marked "YES", or a response to either of these questions is missing.

#### AE Time Since First Dose (Days)

If AE start date < Date of first dose of study treatment then</li>

Time since first dose = AE start date - Date of first dose of study treatment

• If AE start date ≥ Date of first dose of study treatment then

Time since first dose = AE start date – Date of first dose of study treatment +1

Missing if AE start date or date of first dose of study treatment is missing.

### AE Duration (Days)

- AE end date AE start date + 1
- Missing if AE start date or end date is missing.

#### **AESIs**

See Section 11.1.1

# 14.5. Appendix 5: Reporting Standards for Missing Data

## 14.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion is defined as completion of the End of Study (Week<br/>12) visit.</li> </ul> |
| | Withdrawn subjects will not be replaced in the study. |
| | <ul> <li>All available data from subjects who were withdrawn from the study will be listed<br/>and all available planned data will be included in summary tables and figures,<br/>unless otherwise specified.</li> </ul> |
| Pre-Screen<br>and Screen<br>Failures | A subject will be assigned a subject number at the time when the informed consent form (ICF) is signed. |
| | <ul> <li>A subject who is assigned a subject number but does not have any screening<br/>procedures at Visit 1 will be considered a pre-screen failure.</li> </ul> |
| | A subject who completes at least one Visit 1 procedure but does not attempt to self-administer a dose of mepolizumab will be considered a screen failure. |

# 14.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>In general, analysis will be performed on all available data and no imputation will<br/>be performed for missing data. However, if there are withdrawals from the study<br/>due to issues pertaining to the use of the autoinjector, a sensitivity analysis of<br/>the primary analysis will be performed. Missing or "not attempted" injection<br/>success assessments following these withdrawals will be imputed as injection<br/>failures i.e. unsuccessful attempts to self-administer mepolizumab in this<br/>sensitivity analysis.</li> </ul> |
| | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument. These data will be indicated by the use of a "blank" in subject listing displays, unless all data for a specific visit are missing in which case the data is excluded from the listing.</li> <li>Data below the limit of quantification (BLQ) is not missing data and must be</li> </ul> |
| | displayed as such and included in all listings and summaries. |
| Outliers | <ul> <li>Any subjects excluded from the summaries and/or statistical analyses because<br/>their values are considered outliers will be documented along with the reason for<br/>exclusion in the CSR.</li> </ul> |

## 14.5.3. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Missing dates will be indicated by the use of a "blank" in subject listing displays. |
| AEs | <ul> <li>No partial dates will be recorded in this study for AEs or SAEs</li> <li>Missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. AEs with completely missing start dates will be considered to start on-treatment (worst case). </li> </ul> |

## 14.5.4. Handling of Missing Time Point for Assessment of Injection Pain

| Element | Reporting Detail |
|---|---|
| Pain Diary | <ul> <li>Missing nominal time point description (Injection, 1 hour or 24 hours) in the pain diary data may occur if the time of injection is corrected during data cleaning and subsequent pain diary assessments fall out of the eDiary defined time window for the pain assessment.</li> <li>Pain diary assessments with missing nominal timepoint will be assigned to the closest nominal timepoint, unless data already exists at that timepoint, and will be included in summary tables.</li> </ul> |

# 14.6. Appendix 6: Values of Potential Clinical Importance

# 14.6.1. Laboratory Values of Potential Clinical Concern

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Age | Clinical Concern Range | |
| | | Category | Low Flag (< x) | High Flag (>x) |
| Hematocrit | Ratio of 1 | 12+ | 0.201 | 0.599 |
| Haemoglobin | G/L | 12+ | 71 | 199 |
| Platelet Count | GI/L | 1+ | 31 | 1499 |
| White Blood Cell Count (WBC) | GI/L | 12+ | 1.1 | |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Age | Clinical Concern Range | |
| | | Category | Low Flag (< x) | High Flag (>x) |
| ALT | U/L | 3-12 | | >143 (and Total<br>Bilirubin >43) |
| | U/L | 13+ | | >239 (and Total<br>Bilirubin >43) |
| Calcium | mmol/L | 3+ | 1.50 | 3.24 |
| Glucose | mmol/L | 1+ | 2.2 | 27.8 |
| Phosphorus, Inorg | mmol/L | 3+ | 0.32 | |
| Potassium | mmol/L | 3+ | 2.8 | 6.5 |
| Sodium | mmol/L | 0+ | 120 | 160 |

| Possible Hy's Law Cases | | | |
|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range |
| ALT, Bilirubin | | | ALT ≥ 3xULN and Bilirubin ≥ 2xULN (>35% direct) |
| ALT, INR | | | ALT ≥ 3xULN and INR > 1.5 |

### NOTES:

• ULN = Upper Limit of Normal.

# 14.7. Appendix 7: Abbreviations & Trade Marks

## 14.7.1. Abbreviations

| Abbreviation | Description |
|--------------|-------------------------------------------------|
| ADA | Anti-drug Antibody |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AESI | Adverse Events of Special Interest |
| A&R | Analysis and Reporting |
| ASE | All Subjects Enrolled |
| BLQ | Below the Limit of Quantification |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CRF | Case Record Form |
| CSR | Clinical Study Report |
| Ctrough | Concentration at the end of the dosing interval |
| CVT | Cardiac, Vascular and Thromboembolic |
| DBF | Database Freeze |
| DOB | Date of Birth |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| GSK | GlaxoSmithKline |
| ICH | International Conference on Harmonisation |
| ICS | Inhaled Corticosteroid |
| IDSL | Integrated Data Standards Library |
| LLQ | Lower Limit of Quantification |
| NQ | Non-quantifiable |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PSAP | Program Safety Analysis Plan |
| RAP | Reporting & Analysis Plan |
| RTF | Rich Text Format |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SC | Subcutaneous |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| SI | System Independent |
| ULN | Upper Limit of Normal |
| VAS | Visual Analogue Scale |
| WBC | White Blood Cell |
#### 14.7.2. Trademarks

| Trademarks of the GlaxoSmithKline |
|-----------------------------------|
| Group of Companies |

NONE

Trademarks not owned by the GlaxoSmithKline Group of Companies

SAS

## 14.8. Appendix 8: List of Data Displays

## 14.8.1. Study Population Tables

| Study Population - Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.1 | ASE | TAB_POP1 | Summary of Study Populations | | SAC |
| 6.2 | ASE | ES6 | Summary of Screen Failures | Include footnote "Note:<br>Inclusion/exclusion criteria include<br>protocol defined continuation criteria." | SAC |
| 6.3 | ASE | NS1 | Summary of Number of Subjects by Country and Site | "Not Treated" column should be added to include subjects who did not receive treatment. | SAC |
| 6.4 | All Subjects | SD1 | Summary of IP Discontinuation | | SAC |
| 6.5 | All Subjects | ES1 | Summary of Subject Disposition | | SAC |
| 6.6 | All Subjects | DV1 | Summary of Important Protocol Deviations | | SAC |
| 6.7 | All Subjects | EX1 | Summary of Exposure to Study Treatment (months) | Categories 1, 2, 3 months Summary statistics for duration of exposure (months) Include footnote: "Note: For the categorical summary, exposure is rounded to the nearest whole month. | SAC |
| 6.8 | All Subjects | TAB_EX1 | Summary of Injection Site by Visit | | SAC |
| 6.9 | All Subjects | DM1 | Summary of Demographic Characteristics | | SAC |
| 6.10 | All Subjects | DM5 | Summary of Race and Racial Combinations | | SAC |
| 6.11 | ASE | DM11 | Summary of Age Ranges | "Not Treated" column should be added to include subjects who did not receive treatment. | SAC |
| 6.12 | All Subjects | TAB_POP2 | Summary of Disease Duration | | SAC |
| 6.13 | All Subjects | TAB_POP3 | Summary of Prior Experience with Self-Injection of Medication | | SAC |

| Study Population - Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.14 | All Subjects | TAB_POP4 | Summary of Baseline Mepolizumab Use | | SAC |
| 6.15 | All Subjects | TAB_POP5 | Summary of Previous Mepolizumab Clinical Trials | | SAC |
| 6.16 | All Subjects | MH4 | Summary of Past Medical Conditions | | SAC |
| 6.17 | All Subjects | MH4 | Summary of Current Medical Conditions | | SAC |
| 6.18 | All Subjects | FH1 | Summary of Family History of Cardiovascular Risk Factors | | SAC |
| 6.19 | All Subjects | SU1 | Summary of Smoking History | Smoking status (current/former/never) only | SAC |

## 14.8.2. Evaluation of Autoinjector

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Evalua | tion of Autoinje | ector - Tables | | | |
| 7.1 | All Subjects | TAB_INJ1 | Summary of the Proportion of Subjects Successfully Able to Self-Administer Injection by Visit – First Attempt Autoinjector with Standard Label + Pictogram | Add footnote: "Note: If a subject has more than one attempt to selfadminister study treatment at a single visit, only the first attempt is included in this summary." | SAC |
| 7.2 | All Subjects | TAB_INJ1 | Summary of the Proportion of Subjects Successfully Able to Self-Administer Injection by Visit – First Attempt Autoinjector with Standard Label | Add footnote: "Note: If a subject has more than one attempt to self-administer study treatment at a single visit, only the first attempt is included in this summary." | SAC |
| 7.3 | All Subjects | TAB_INJ1 | Summary of the Proportion of Subjects Successfully Able to Self-Administer Injection by Visit – Best Attempt Autoinjector with Standard Label + Pictogram | Add footnote: "Note: If a subject has more than one attempt to self-administer study treatment at a single visit, the best attempt is included in this summary." | SAC |
| 7.4 | All Subjects | TAB_INJ1 | Summary of the Proportion of Subjects Successfully Able to Self-Administer Injection by Visit – Best Attempt Autoinjector with Standard Label | Add footnote: "Note: If a subject has more than one attempt to self-administer study treatment at a single visit, the best attempt is included in this summary." | SAC |
| 7.5 | All Subjects | TAB_INJ2 | Summary of Investigator Evaluation of User/Device Errors by Visit Autoinjector with Standard Label + Pictogram | Add footnote: "Note: If a subject has more than one attempt to self-administer study treatment at a single visit, only the first attempt is included in this summary." | SAC |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Evaluat | tion of Autoinje | ector - Tables | | , | |
| 7.6 | All Subjects | TAB_INJ2 | Summary of Investigator Evaluation of User/Device Errors by Visit Autoinjector with Standard Label | Add footnote: "Note: If a subject has more than one attempt to self-administer study treatment at a single visit, only the first attempt is included in this summary." | SAC |
| 7.7 | All Subjects | TAB_INJ3 | Summary of Observer Checklist for In-Clinic Injections Autoinjector with Standard Label + Pictogram | Add footnote: "Note: If a subject has more than one attempt to self-administer study treatment at a single visit, only the first attempt is included in this summary." | SAC |
| 7.8 | All Subjects | TAB_INJ3 | Summary of Observer Checklist for In-Clinic Injections Autoinjector with Standard Label | Add footnote: "Note: If a subject has more than one attempt to self-administer study treatment at a single visit, only the first attempt is included in this summary." | SAC |
| 7.9 | All Subjects | TAB_INJ4 | Summary of Subject Completed Checklist for At-Home Injection at Week 4 Autoinjector with Standard Label + Pictogram | Add footnote: "Note: If a subject has more than one attempt to self-administer study treatment at a single visit, only the first attempt is included in this summary." | SAC |
| 7.10 | All Subjects | TAB_INJ4 | Summary of Subject Completed Checklist for At-Home Injection at Week 4 Autoinjector with Standard Label | Add footnote: "Note: If a subject has more than one attempt to self-administer study treatment at a single visit, only the first attempt is included in this summary." | SAC |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Evaluat | ion of Autoinje | ector - Tables | | | |
| 7.11 | All Subjects | TAB_INJ5 | Summary of Device Usability/Functionality Questionnaire Autoinjector with Standard Label + Pictogram | Add footnote: "Note: Questionnaire was not completed by subjects who took part in liquid safety syringe study 205667." | SAC |
| 7.12 | All Subjects | TAB_INJ5 | Summary of Device Usability/Functionality Questionnaire Autoinjector with Standard Label | Add footnote: "Note: Questionnaire was not completed by subjects who took part in liquid safety syringe study 205667." | SAC |
| 7.13 | All Subjects | LIST_INJ1 | Listing of Investigator Assessment of Injection Success -<br>Subjects Requiring More Than One Attempt to Self-Administer<br>Mepolizumab at any Visit | Include treatment and label description in by-line. | SAC |

### 14.8.3. Pharmacokinetic Analyses

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| PK Concentration: Figures | | | | | |
| 8.1 | PK | PK16a | Individual Plasma Mepolizumab Concentration-Time Plots (Linear and Semi-Log) by Subject | Subject number and baseline mepolizumab use as by-line. Indicate the injection site used for each dose using different plotting characters. | SAC |
| 8.2 | PK | PK26 | Individual Plasma Mepolizumab Concentration-Time Plots (Linear and Semi-Log) by Baseline Mepolizumab Use | Baseline mepolizumab use as a by-line. All subjects in the same baseline mepolizumab group on the same graph ("spaghetti" plot). Due to the number of subjects, legend to identify subjects is not required. | SAC |
| 8.3 | PK | PK26 | Individual Plasma Mepolizumab Concentration-Time Plots (Linear and Semi-Log) by Baseline Mepolizumab Use and Injection Site – Subjects Using the Same Injection Site Throughout the Study | Baseline mepolizumab use and injection site as a by-line. All subjects in the same baseline mepolizumab group and injection site on the same graph ("spaghetti" plot). Include only the subset of subjects using the same injection site for all doses of study treatment. Due to the number of subjects, legend to identify subjects is not required. | SAC |
| 8.4 | PK | PK19 | Mean Plasma Mepolizumab Concentration-Time Plots by Baseline Mepolizumab Use (Linear and Semi-Log) | Include (N=XX) in legend. | SAC |
| 8.5 | PK | PK18 | Median Plasma Mepolizumab Concentration-Time Plots by Baseline Mepolizumab Use (Linear and Semi-Log) | Include (N=XX) in legend. | SAC |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 8.6 | PK | PK19 | Mean Plasma Mepolizumab Concentration-Time Plots by<br>Baseline Mepolizumab Use and Injection Site (Linear and Semi-<br>Log) – Subjects Using the Same Injection Site Throughout the<br>Study | Include only the subset of subjects using the same injection site for all doses of study treatment. Include (N=XX) in legend. | SAC |
| 8.7 | PK | PK18 | Median Plasma Mepolizumab Concentration-Time Plots by Baseline Mepolizumab Use and Injection Site (Linear and Semi-Log) – Subjects Using the Same Injection Site Throughout the Study | Include only the subset of subjects using the same injection site for all doses of study treatment. Include (N=XX) in legend. | SAC |
| 8.8 | PK | - | Scatter Plot of Individual Plasma Mepolizumab Concentration-<br>Time Data by Week 12 Binding Antibody Result | Use grey open circles for data points for subjects with negative binding antibody. Use larger filled blue circles for data points for subjects with positive binding antibody, and annotate data points with subject number. | SAC |
| Pharma | cokinetic – Ta | bles | | | |
| 8.1 | PK | PK01 | Summary of Plasma Mepolizumab Concentration-Time Data | | SAC |
| 8.2 | PK | PK01 | Summary of Plasma Mepolizumab Concentration-Time Data by Baseline Mepolizumab Use | | SAC |
| 8.3 | PK | PK01 | Summary of Plasma Mepolizumab Concentration-Time Data by Baseline Mepolizumab Use and Injection Site – Subjects Using the Same Injection Site Throughout the Study | Include only the subset of subjects using the same injection site for all doses of study treatment. | SAC |

## 14.8.4. Pharmacodynamic Analyses

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Pharma | harmacodynamic – Figures | | | | |
| 9.1 | PD | FIG_PD1 | Geometric Mean (95% CI) Absolute Blood Eosinophils by Visit and Baseline Mepolizumab Use | Include (N=XX) in legend. | SAC |
| 9.2 | PD | FIG_PD1 | Geometric Mean (95% CI) Absolute Blood Eosinophils by Visit,<br>Baseline Mepolizumab Use and Injection Site – Subjects Using<br>the Same Injection Site Throughout the Study | Baseline mepolizumab use as by-line. Separate lines on graph corresponding to injection sites. Include only the subset of subjects using the same injection site for all doses of study treatment. Include (N=XX) in legend. | SAC |
| 9.3 | PD | FIG_PD1 | Geometric Mean (95% CI) Ratio to Baseline Blood Eosinophils by Visit and Baseline Mepolizumab Use | Include (N=XX) in legend. | SAC |
| 9.4 | PD | FIG_PD1 | Geometric Mean (95% CI) Ratio to Baseline Blood Eosinophils by Visit, Baseline Mepolizumab Use and Injection Site – Subjects Using the Same Injection Site Throughout the Study | Baseline mepolizumab use as by-line. Separate lines on graph corresponding to injection sites. Include only the subset of subjects using the same injection site for all doses of study treatment. Include (N=XX) in legend. | SAC |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 9.5 | PD | - | Scatter Plot of Individual Blood Eosinophil-Time Data by Week 12 Binding Antibody Result | Use grey open circles for data points for subjects with negative binding antibody. Use larger filled blue circles for data points for subjects with positive binding antibody, and annotate data points with subject number. | SAC |
| Pharma | codynamic – T | ables | | | |
| 9.1 | PD | TAB_PD1 | Summary of Blood Eosinophils (Gl/L) by Visit | | SAC |
| 9.2 | PD | TAB_PD2 | Summary of Ratio to Baseline Blood Eosinophils by Visit | | SAC |
| 9.3 | PD | TAB_PD3 | Summary of Blood Eosinophils by Visit and Baseline<br>Mepolizumab Use | | SAC |
| 9.4 | PD | TAB_PD4 | Summary of Ratio to Baseline Blood Eosinophils by Visit and Baseline Mepolizumab Use | | SAC |
| 9.5 | PD | TAB_PD3 | Summary of Blood Eosinophils by Visit, Baseline Mepolizumab<br>Use and Injection Site– Subjects Using the Same Injection Site<br>Throughout the Study | Add baseline mepolizumab use to by line, and include injection site in first column. Include only the subset of subjects using the same injection site for all doses of study treatment. | SAC |
| 9.6 | PD | TAB_PD4 | Summary of Ratio to Baseline Blood Eosinophils by Visit,<br>Baseline Mepolizumab Use and Injection Site– Subjects Using<br>the Same Injection Site Throughout the Study | Add baseline mepolizumab use to by line, and include injection site in first column. Include only the subset of subjects using the same injection site for all doses of study treatment. | SAC |

#### 14.8.5. Exacerbations

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Exacert | Exacerbations: Tables | | | | |
| 10.1 | All Subjects | TAB_EX1 | Summary of Number of Subjects with at Least One On-Treatment Exacerbation | | SAC |

## 14.8.6. Safety Analyses

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Safety : | Figures | | | | |
| Advers | e Events | | | | |
| 11.1 | All Subjects | LIVER14 | Scatter Plot of Maximum vs Baseline for ALT | If there are unscheduled assessments add footnote: "Note: Maximum Value includes scheduled and unscheduled assessments." | SAC |
| 11.2 | All Subjects | LIVER9 | Scatter Plot of Maximum Total Bilirubin vs Maximum ALT | If there are unscheduled assessments add footnote: "Note: Maximum Value includes scheduled and unscheduled assessments." | SAC |
| Safety : | Tables | | | | |
| Advers | e Events | | | | |
| 11.1 | All Subjects | AE1 | Summary of All On-Treatment Adverse Events by System Organ Class and Preferred Term | | SAC |
| 11.2 | All Subjects | AE1 | Summary of All Post-Treatment Adverse Events by System<br>Organ Class and Preferred Term | | SAC |
| 11.3 | All Subjects | AE3 | Summary of Common (>=3% Incidence) On-Treatment Adverse Events by Overall Frequency | | SAC |
| 11.4 | All Subjects | AE15 | Summary of Common (>=3% Incidence) On-Treatment Non-<br>Serious Adverse Events by System Organ Class and Preferred<br>Term (Number of Subjects and Occurrences) | | SAC |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Safety : | Figures | | | | · |
| 11.5 | All Subjects | AE5A | Summary of All On-Treatment Adverse Events by Maximum Intensity by System Organ Class and Preferred Term | | SAC |
| 11.6 | All Subjects | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term | | SAC |
| 11.7 | All Subjects | AE5A | Summary of All Drug-Related Adverse Events by Maximum Intensity by System Organ Class and Preferred Term | | SAC |
| 11.8 | All Subjects | AE1 | Summary of On-Treatment Adverse Events by Week 12 Binding Antibody Result | Add in row with n in each binding antibody result category. See Section 12. | SAC |
| 11.9 | All Subjects | AE3 | Summary of All Adverse Events Leading to Permanent Discontinuation from Study Treatment and/or Withdrawal from the Study by Overall Frequency | | SAC |
| 11.10 | All Subjects | AE1 | Summary of Adverse Events Reported on the Day of Dosing by System Organ Class and Preferred Term | | SAC |
| 11.11 | All Subjects | AE7 | Listing of Subject Numbers for Individual On-Treatment Adverse Events | | SAC |
| 11.12 | All Subjects | AE2 | Listing of Relationship of Adverse Event, System Organ Classes, Preferred Terms and Verbatim Text | | SAC |
| Serious | Adverse Even | ts | | | |
| 11.13 | All Subjects | AE3 | Summary of Fatal Serious Adverse Events by Overall Frequency | | SAC |
| 11.14 | All Subjects | AE3 | Summary of Drug-Related Fatal Serious Adverse Events by<br>Overall Frequency | | SAC |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Safety | Figures | | | | |
| 11.15 | All Subjects | AE1 | Summary of All On-Treatment Serious Adverse Events by System Organ Class and Preferred Term | | SAC |
| 11.16 | All Subjects | AE16 | Summary of All On-Treatment Serious Adverse Events by<br>System Organ Class and Preferred Term (Number of Subjects<br>and Occurrences) | | SAC |
| 11.17 | All Subjects | AE1 | Summary of All Post-Treatment Serious Adverse Events by System Organ Class and Preferred Term | | SAC |
| 11.18 | All Subjects | AE1 | Summary of All Pre-Treatment Serious Adverse Events by System Organ Class and Preferred Term | | SAC |
| 11.19 | All Subjects | AE1 | Summary of All Drug-Related Serious Adverse Events by<br>System Organ Class and Preferred Term | | SAC |
| Advers | e Events of Sp | ecial Interest | | 1 | |
| 11.20 | All Subjects | AE1 | Summary of On-Treatment Adverse Events Reported by the Investigator as Meeting the Criteria for Anaphylaxis | | SAC |
| 11.21 | All Subjects | TAB_S1 | Summary Profile of On-Treatment Adverse Events Reported by the Investigator as Meeting the Criteria for Anaphylaxis | | SAC |
| 11.22 | All Subjects | AE1 | Summary of On-Treatment Adverse Events Defined by the Investigator as Systemic Reactions - Allergic (Type I Hypersensitivity) and Other Systemic | | SAC |
| 11.23 | All Subjects | TAB_S1 | Summary Profile of On-Treatment Adverse Events Defined by the Investigator as Systemic Reactions - Allergic (Type I Hypersensitivity) and Other Systemic | | SAC |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Safety : | Figures | | | | |
| 11.24 | All Subjects | AE1 | Summary of On-Treatment Adverse Events Defined by the Investigator as Systemic Reactions - Allergic (Type I Hypersensitivity) | | SAC |
| 11.25 | All Subjects | TAB_S1 | Summary Profile of On-Treatment Adverse Events Defined by the Investigator as Systemic Reactions - Allergic (Type I Hypersensitivity) | | SAC |
| 11.26 | All Subjects | AE1 | Summary of On-Treatment Adverse Events Defined by the Investigator as Systemic Reactions – Other Systemic | | SAC |
| 11.27 | All Subjects | TAB_S1 | Summary Profile of On-Treatment Adverse Events Defined by the Investigator as Systemic Reactions - Other Systemic | | SAC |
| 11.28 | All Subjects | AE1 | Summary of On-Treatment Adverse Events Defined by the Investigator as Local Injection Site Reactions | | SAC |
| 11.29 | All Subjects | TAB_S1 | Summary Profile of On-Treatment Adverse Events Defined by the Investigator as Local Injection Site Reactions | | SAC |
| 11.30 | All Subjects | AE1 | Summary of On-Treatment Adverse Events Categorised as Serious Cardiac, Vascular and Thromboembolic Events | | SAC |
| 11.31 | All Subjects | TAB_S1 | Summary Profile of On-Treatment Adverse Events Categorised as Serious Cardiac, Vascular and Thromboembolic Events | | SAC |
| 11.32 | All Subjects | AE1 | Summary of On-Treatment Adverse Events Categorised as Serious Ischemic Events | | SAC |
| 11.33 | All Subjects | TAB_S1 | Summary Profile of On-Treatment Adverse Events Categorised as Serious Ischemic Events | | SAC |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Safety : | Safety : Figures | | | | |
| 11.34 | All Subjects | AE1 | Summary of On-Treatment Adverse Events Categorised as Malignancies | | SAC |
| 11.35 | All Subjects | TAB_S1 | Summary Profile of On-Treatment Adverse Events Categorised as Malignancies | | SAC |
| 11.36 | All Subjects | AE1 | Summary of On-Treatment Adverse Events Categorised as Opportunistic Infections | | SAC |
| 11.37 | All Subjects | TAB_S1 | Summary Profile of On-Treatment Adverse Events Categorised as Opportunistic Infections | | SAC |
| Labora | tory - Haemato | logy | | | |
| 11.38 | All Subjects | LB1 | Summary of Haematology Changes from Baseline by Visit | Include baseline values | SAC |
| 11.39 | All Subjects | LB3 | Summary of Haematology Shifts from Baseline Relative to Normal Range by Visit | | SAC |
| 11.40 | All Subjects | LB3 | Summary of Haematology Shifts from Baseline Relative to PCI Criteria by Visit | | SAC |
| Labora | tory – Clinical ( | Chemistry | | | |
| 11.41 | All Subjects | LB1 | Summary of Clinical Chemistry Changes from Baseline by Visit | Include baseline values | SAC |
| 11.42 | All Subjects | LB3 | Summary of Clinical Chemistry Shifts from Baseline Relative to Normal Range by Visit | | SAC |
| 11.43 | All Subjects | LB3 | Summary of Clinical Chemistry Shifts from Baseline Relative to PCI Criteria by Visit | | SAC |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Safety : | Safety : Figures | | | | |
| ECG | | | | | |
| 11.43 | All Subjects | EG1 | Summary of ECG Findings by Visit | | SAC |
| 11.45 | All Subjects | EG2 | Summary of ECG Values by Visit | | SAC |
| 11.46 | All Subjects | EG2 | Summary of Change from Baseline in ECG Values by Visit | Include baseline values | SAC |
| 11.47 | All Subjects | TAB_ECG1 | Summary of Actual and Change From Baseline QTc(F) Values by Category (msec) | If there are unscheduled ECGs, include<br>"Maximum Value Post Baseline" as an<br>additional timepoint and add footnote:<br>"Note: Maximum Value Post-Baseline<br>includes scheduled and unscheduled<br>assessments." | SAC |
| 11.48 | All Subjects | TAB_ECG1 | Summary of Actual and Change From Baseline QTc(B) Values by Category (msec) | If there are unscheduled ECGs, include "Maximum Value Post Baseline" as an additional timepoint and add footnote: "Note: Maximum Value Post-Baseline includes scheduled and unscheduled assessments." | SAC |
| 11.49 | All Subjects | TAB_ECG1 | Summary of Actual and Change From Baseline QTc (Correction Unspecified) Values by Category (msec) | If there are unscheduled ECGs, include "Maximum Value Post Baseline" as an additional timepoint and add footnote: "Note: Maximum Value Post-Baseline includes scheduled and unscheduled assessments." | SAC |
| Vital Sig | gns | | | | |
| 11.50 | All Subjects | VS1 | Summary of Vital Signs by Visit | | SAC |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Safety : | Safety : Figures | | | | |
| 11.51 | All Subjects | VS1 | Summary of Change from Baseline in Vital Signs by Visit | Include baseline values | SAC |
| Injectio | n Pain Assessı | ments | | | |
| 11.52 | All Subjects | TAB_S3 | Summary of Injection Pain – VAS Scores (mm) | By Visit and time point post-injection (injection, 1 hr post, 24 hrs post) | SAC |
| 11.53 | All Subjects | TAB_S4 | Summary of Injection Pain – Categorical Pain Assessment | By Visit and time point post-injection (injection, 1 hr post, 24 hrs post) | SAC |

## 14.8.7. Immunogenicity

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Immun | nmunogenicity : Tables | | | | |
| 12.1 | All Subjects | TAB_S2 | Summary of Binding Antibody by Visit | Positive/Negative at Week 0 and Week 12/Early Withdrawal. For Week 12/Early Withdrawal, include min, median, max values for titre. | SAC |
| 12.2 | All Subjects | TAB_S2 | Summary of Binding Antibody by Visit and Baseline<br>Mepolizumab Use | Positive/Negative at Week 0 and Week 12/Early Withdrawal. For Week 12/Early Withdrawal, include min, median, max values for titre. | SAC |
| 12.3 | All Subjects | TAB_S2 | Summary of Binding Antibody – Subjects Without Positive Result at Week 0 | Positive/Negative at Week 12/Early<br>Withdrawal, include min, median, max<br>values for titre. | SAC |
| 12.4 | All Subjects | TAB_S2 | Summary of Neutralising Antibody by Visit | No titre values available for Neutralising antibody. | SAC |
| 12.5 | All Subjects | TAB_S2 | Summary of Neutralising Antibody by Visit and Baseline Mepolizumab Use | No titre values available for Neutralising antibody. | SAC |

## 14.8.8. ICH and Other Listings

| | | IDSL / TST ID | | | |
|---|---|---|---|---|---|
| No. | Population | / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study | Population | 1 | | | |
| 1 | ASE | ES7 | Listing of Reasons for Screen Failure | Include footnote "Note:<br>Inclusion/exclusion criteria include<br>protocol defined continuation criteria." | SAC |
| 2 | All Subjects | SP3 | Listing of Subjects Excluded from Any Population | | SAC |
| 3 | All Subjects | SD2 | Listing of Reasons for Study Treatment Discontinuation | | SAC |
| 4 | All Subjects | ES2 | Listing of Reasons for Study Withdrawal | | SAC |
| 5 | All Subjects | DV2 | Listing of Important Protocol Deviations | | SAC |
| 6 | All Subjects | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | Include any deviations in protocol defined continuation criteria. | SAC |
| 7 | All Subjects | EX3 | Listing of Exposure Data | Include the following additional variables: injection site, investigator assessment of injection success. Include treatment and label description. | SAC |
| 8 | All Subjects | LIST_INJ2 | Listing of Person Administering Injection[1] and Time From Removal of Autoinjector from Storage to Injection | Include data for all 3 doses. Footnote: "[1] For the at-home injection (week 4), the person administering the injection is documented by the eDiary as the user (caregiver/patient) who logged in to complete the at-home injection checklist." | SAC |

| ICH an | ICH and Other Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 9 | All Subjects | DM2 | Listing of Demographic Characteristics | | SAC |
| 10 | All Subjects | DM9 | Listing of Race | | SAC |
| 11 | All Subjects | LIST_POP1 | Listing of Baseline Mepolizumab Use | | SAC |
| 12 | All Subjects | LIST_POP2 | Listing of Previous Mepolizumab Clinical Trials | | SAC |
| 13 | All Subjects | MH2 | Listing of Medical Conditions | | SAC |
| 14 | All Subjects | FH5 | Listing of Family History | | SAC |
| 15 | All Subjects | CM3 | Listing of Concomitant Medications | Include all data collected on the CRF, plus study day for start date | |
| Evalua | tion of Autoinjector | • | | | |
| 16 | All Subjects | LIST_INJ1 | Listing of Investigator Assessment of Injection Success | Include treatment and label description in by-line. | SAC |
| 17 | All Subjects | - | Listing of Observer Checklist for In-Clinic Injections | Include treatment and label description in by-line. Exclude information presented in Listing 8. | SAC |
| 18 | All Subjects | - | Listing of Subject Completed Checklist for At-Home Injection at Week 4 | Include treatment and label description in by-line. Exclude information presented in Listing 8. | SAC |
| 19 | All Subjects | - | Listing of Device Usability/Functionality Questionnaire | Include treatment and label description in by-line. | SAC |

| ICH an | d Other Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Co | ncentration | 1 | | | |
| 20 | PK | PK07 | Listing of Plasma Concentration-Time Data | | SAC |
| Exacei | bations | | | · | |
| 21 | All Subjects | LIST_EX1 | Listing of Exacerbations | | SAC |
| Advers | se Events | | | · | |
| 22 | All Subjects | AE8 | Listing of All Adverse Events | Add phase: Pre-treatment, on-treatment, post-treatment (see Section 14.2.1.1). Include treatment in by-line. | SAC |
| 23 | All Subjects | AE8 | Listing of Adverse Events Leading to Withdrawal From Study | Add phase: Pre-treatment, on-treatment, post-treatment (see Section 14.2.1.1). Include treatment in by-line. | SAC |
| 24 | All Subjects | AE8 | Listing of Adverse Events Reported on the Day of Dosing | Add phase: Pre-treatment, on-treatment, post-treatment (see Section 14.2.1.1). Include treatment in by-line. | SAC |
| Seriou | s Adverse Events | • | | | |
| 25 | All Subjects | AE8 | Listing of Fatal Serious Adverse Events | Add phase: Pre-treatment, on-treatment, post-treatment (see Section 14.2.1.1). Include treatment in by-line. | SAC |

| ICH an | d Other Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 26 | All Subjects | AE8 | Listing of Non-Fatal Serious Adverse Events | Add phase: Pre-treatment, on-treatment, post-treatment (see Section 14.2.1.1). Include treatment in by-line. | SAC |
| 27 | All Subjects | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | Include treatment in by-line. | SAC |
| Advers | se Events of Special | Interest | | | |
| 28 | All Subjects | AE8 | Listing of Adverse Events Reported by the Investigator as Meeting the Criteria for Anaphylaxis | Add phase: Pre-treatment, on-treatment, post-treatment (see Section 14.2.1.1). Add injection reaction symptoms and number of doses prior to event. Include treatment in by-line. | SAC |
| 29 | All Subjects | AE8 | Listing of Adverse Events Defined by the Investigator as Systemic Reactions - Allergic (Type I Hypersensitivity) | Add phase: Pre-treatment, on-treatment, post-treatment (see Section 14.2.1.1). Add injection reaction symptoms and number of doses prior to event. Include treatment in by-line. | SAC |
| 30 | All Subjects | AE8 | Listing of Adverse Events Defined by the Investigator as Systemic Reactions – Other Systemic | Add phase: Pre-treatment, on-treatment, post-treatment (see Section 14.2.1.1). Add injection reaction symptoms and number of doses prior to event. Include treatment in by-line. | SAC |

| ICH an | ICH and Other Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 31 | All Subjects | AE8 | Listing of Adverse Events Defined by the Investigator as Local Injection Site Reactions | Add phase: Pre-treatment, on-treatment, post-treatment (see Section 14.2.1.1). Add injection reaction symptoms and number of doses prior to event. Include treatment in by-line. | SAC |
| 32 | All Subjects | AE8 | Listing of Adverse Events Categorised as Serious Cardiac,<br>Vascular and Thromboembolic Events | Add phase: Pre-treatment, on-treatment, post-treatment (see Section 14.2.1.1). Include treatment in by-line. | SAC |
| 33 | All Subjects | AE8 | Listing of Adverse Events Categorised as Serious Ischemic Events | Add phase: Pre-treatment, on-treatment, post-treatment (see Section 14.2.1.1). Include treatment in by-line. | SAC |
| 34 | All Subjects | AE8 | Listing of Adverse Events Categorised as Malignancies | Add phase: Pre-treatment, on-treatment, post-treatment (see Section 14.2.1.1). Include treatment in by-line. | SAC |
| 35 | All Subjects | AE8 | Listing of Adverse Events Categorised as Opportunistic Infections | Add phase: Pre-treatment, on-<br>treatment, post-treatment (see Section<br>14.2.1.1).<br>Include treatment in by-line. | SAC |

| ICH and Other Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | atory | | | | |
| 36 | All Subjects | LB5 | Listing of Haematology Data for Subjects with Abnormalities of Potential Clinical Concern | Include treatment in by-line. | SAC |
| 37 | All Subjects | LB5 | Listing of Chemistry Data for Subjects with Abnormalities of Potential Clinical Concern | Include treatment in by-line. | SAC |
| ECG | | | | | |
| 38 | All Subjects | EG3 | Listing of ECG Values (Subjects with QTc >500 msec or Increase >= 60 msec from Baseline) | Include treatment in by-line. | SAC |
| Injecti | on Pain | | | | |
| 39 | All Subjects | LIST_S1 | Listing of Injection Pain Assessment | Include treatment in by-line. | SAC |
| Immunogenicity | | | | | |
| 40 | All Subjects | IMM2 | Listing of Immunogenicity Data for Subjects with at Least One Positive Screening Binding Assay | Include columns for Screening Binding<br>Assay, Confirmation Binding Assay,<br>Confirmation Binding Assay Titre,<br>Transient/Persistent, Neutralising<br>Antibody Assay | SAC |
| PD | | | | | |
| 41 | Pharmacodynamic | LIST_PD1 | Listing of Blood Eosinophils | | SAC |

#### 14.9. Appendix 9: Example Mock Shells for Data Displays

Example TAB\_POP1 Protocol: 204959

Population: All Subjects Enrolled


# Table X Summary of Study Populations

| Population | Liquid Autoinjector (N=XX) |
|----------------------------------------------|----------------------------|
| All Subjects Enrolled | XX |
| All Subjects (Safety) | XX (XX%) |
| Autoinjector with Standard Label + Pictogram | XX (XX%) |
| Autoinjector with Standard Label | XX (XX%) |
| Pharmacokinetic | XX (XX%) |
| Pharmacodynamic | XX (XX%) |

204959


Liquid Autoinjector

Example TAB\_POP2 Protocol: 204959

Population: All Subjects (Safety)

Table X
Summary of Disease Duration

| | | (N=XX) |
|-----------------------------|------------|----------|
| Duration of Disease (years) | n | XX |
| | >=1 to <5 | XX (XX%) |
| | >=5 to <10 | XX (XX%) |
| | etc. | XX (XX%) |
| | Mean | XX.X |
| | SD | XX.XX |
| | Median | XX.X |
| | Minimum | XX |
| | Maximum | XX |

204959


Example TAB\_EX1
Protocol: 204959

Population: All Subjects (Safety)

# Table X Summary of Injection Site

| Visit | Injection Site | Liquid Autoinjector (N=XX) |
|--------|---------------------------------|----------------------------|
| WEEK 0 | n | XX |
| | Abdomen | XX (XX%) |
| | Upper arm | XX (XX%) |
| | Thigh | XX (XX%) |
| | Other, or intervention required | XX (XX%) |
| WEEK 4 | n | XX |
| | Abdomen | XX (XX%) |
| | Upper arm | XX (XX%) |
| | Thigh | XX (XX%) |
| | Other | XX (XX%) |
| WEEK 8 | n | XX |
| WEEK 0 | Abdomen | XX (XX%) |
| | Upper arm | XX (XX%) |
| | Thigh | XX (XX%) |
| | Other, or intervention required | XX (XX%) |

204959

Example TAB\_POP3 Protocol: 204959

Protocol: 204959 

Population: All Subjects (Safety)

| | Liquid Autoinjector (N=XX) |
|---|---|
| n | XX |
| No | XX (XX%) |
| Yes | XX (XX%) |
| Autoinjector (Pen) | XX (XX%) |
| Prefilled syringe | XX (XX%) |
| Vial and syringe | XX (XX%) |
| Other method | XX (XX%) |
| | No Yes Autoinjector (Pen) Prefilled syringe Vial and syringe |


Example TAB\_POP4 Protocol: 204959

Population: All Subjects (Safety)

Table X
Summary of Baseline Mepolizumab Use

| | | Liquid Autoinjector<br>(N=XX) |
|---|---|---|
| Is the subject currently receiving treatment with mepolizumab? | n | XX |
| | No | XX (XX%) |
| | Yes | XX (XX%) |
| Blood eosinophil count criteria met [1][2]? | n | |
| | No | XX (XX%) |
| | Yes | XX (XX%) |
| Most recent blood eosinophil count prior to starting mepolizumab (cells/uL) [2] | n | xx |
| | Median | XX.X |
| | Minimum | XX |
| | Maximum | XX |

<sup>[1]</sup> Blood eosinophil count immediately before starting mepolizumab that was  $\geq$ = 150 cells/uL or a blood eosinophil count that was  $\geq$ = 300 cells/uL in the 12 months prior to starting mepolizumab.

<sup>[2]</sup> Subjects currently receiving treatment with mepolizumab only.

204959


Example TAB\_POP5 Protocol: 204959

Population: All Subjects (Safety)

Table X
Summary of Previous Mepolizumab Clinical Trials

| | | Liquid Autoinjector (N=XX) |
|---|---|---|
| Did the subject participate in a previous mepolizumab trial? | n | XX |
| | No | XX (XX%) |
| | Yes | XX (XX%) |
| Protocol number | 115666 | XX (XX%) |
| | 204471 | XX (XX%) |
| | 205667 | XX (XX%) |

Example TAB\_INJ1

Protocol: 204959 

Population: All Subjects (Safety)

Table X

Summary of Proportion of Subjects Successfully Able to Self-Administer Injection by Visit - First Attempt

Autoinjector with Standard Label + Pictogram

| | Liquid Autoinjector $(N = XX)$ | |
|---|---|---|
| | Attempted Injections | Successful Injections [1] |
| Visit | n (%) | n (%) 95% CI |
| WEEK 0 | XX (XX%) | XX (XX%) (XX%, XX%) |
| WEEK 4 | XX (XX%) | XX (XX%) (XX%, XX%) |
| WEEK 8 | XX (XX%) | XX (XX%) (XX%, XX%) |
| WEEK 4 and 8 | XX (XX%) | XX (XX%) (XX%, XX%) |
| WEEK 0, 4 and 8 | XX (XX%) | XX (XX%) (XX%, XX%) |

[1] The denominator for the percentage of successful injections is the number of attempted injections.

Note: If a subject has more than one attempt to self-administer study treatment at a single visit, only the first attempt is included in this summary.


Example TAB\_INJ2 Protocol: 204959

Population: All Subjects (Safety)

# Table X.X Summary of Investigator Evaluation of User/Device Errors by Visit Autoinjector with Standard Label + Pictogram

| Visit | n | | | Liqu | id Autoinjector (N=XX) |
|---|---|---|---|---|---|
| WEEK 0 | XX | Was the drug successfully injected? | Yes | XX | (XX%) |
| | | 5 | No | XX | (XX%) |
| | | | Not attempted | XX | (XX%) |
| | | User Error | Any User Error | XX | (XX%) |
| | | | Ring cap not removed from autoinjector | XX | (XX%) |
| | | | Autoinjector not properly activated on injection site (e.g., gold needle guard not flush with skin) | | (XX%) |
| | | | Autoinjector used upside down | XX | (XX%) |
| | | | Autoinjector pulled away before end of injection (i.e., before purple indicator stopped moving) | | (XX%) |
| | | | Other | XX | (XX%) |
| | | Device Error | Any Device Error | XX | (XX%) |
| | | | Autoinjector leaking | XX | (XX%) |
| | | | Components missing / broken / cracked | XX | (XX%) |
| | | | Inspection window not clear | XX | (XX%) |
| | | | Cannot remove ring cap | XX | (XX%) |
| | | | Bent needle | XX | (XX%) |
| | | | Cannot push the gold needle guard down to activate (i.e., force too high) | XX | (XX%) |
| | | | Autoinjector does not activate (after pressing gold needle guard down) | XX | (XX%) |

Note: If a subject has more than one attempt to self-administer study treatment at a single visit, only the first attempt is included in this summary.

userid: /arenv/arprod/compound/study/final/drivers/drivername.sas DDMMMYYYY HH:MM Programming Note: Continue for Week 4 and 8

204959


Liquid Autoinjector

Example TAB\_INJ3
Protocol: 204959

Population: All Subjects (Safety)

-

# Table X.X Summary of Observer Checklist for In-Clinic Injections Autoinjector with Standard Label + Pictogram

Visit: WEEK 0

| | | (N=XX) |
|---|---|---|
| Time from removal of pen from storage to injection (mins) | n | XX |
| | Mean | XX.X |
| | SD | XX.XX |
| | Median | XX.X |
| | Minimum | XX |
| | Maximum | XX |
| Confirm who will be administering the injection | n | XX |
| | Patient | XX (XX%) |
| | Caregiver | XX (XX%) |
| Subject/caregiver completed all the training required | n | XX |
| | Yes | XX (XX%) |
| | No | XX (XX%) |
| Subject/caregiver had instructions for use (IFU) available for review | n | XX |
| during injection (as recommended) | | |
| | Yes | XX (XX%) |
| | No | XX (XX%) |

<sup>[1]</sup> Subject / caregiver completed task easily without repeated reference to the IFU.

Note: If a subject has more than one attempt to self-administer study treatment at a single visit, only the first attempt is included in this summary.

<sup>[2]</sup> Subject / caregiver completed task but with some difficulty or repeated reference to the IFU for assistance.

<sup>[3]</sup> Subject / caregiver was not able to (or did not) complete task after multiple attempts and reference to the IFU, or intervention was required.

204959


Liquid Autoinjector

Example TAB\_INJ3 (cont.)

Protocol: 204959

Population: All Subjects (Safety)

Table X.X
Summary of Observer Checklist for In-Clinic Injections
Autoinjector with Standard Label + Pictogram

Visit: WEEK 0

| | | (N=XX) |
|---|---|---|
| Check that the subject / caregiver looks at the label to check the expiration date on the pen prior to use. | n | XX |
| | Easily [1] | XX (XX%) |
| | With some difficulty [2] | XX (XX%) |
| | Did not complete [3] | XX (XX%) |
| Check that the subject / caregiver looks in the inspection window to check the liquid prior to use. | n | XX |
| | Easily [1] | XX (XX%) |
| | With some difficulty [2] | XX (XX%) |
| | Did not complete [3] | XX (XX%) |

- [1] Subject / caregiver completed task easily without repeated reference to the IFU.
- [2] Subject / caregiver completed task but with some difficulty or repeated reference to the IFU for assistance.
- [3] Subject / caregiver was not able to (or did not) complete task after multiple attempts and reference to the IFU, or intervention was required.

Note: If a subject has more than one attempt to self-administer study treatment at a single visit, only the first attempt is included in this summary.
204959

Example TAB\_INJ3 (cont.)

Protocol: 204959

Population: All Subjects (Safety)


# Table X.X Summary of Observer Checklist for In-Clinic Injections Autoinjector with Standard Label + Pictogram

Visit: WEEK 0

| | | Liquid Autoinjector (N=XX) |
|---|---|---|
| Check that the subject / caregiver removes the clear needle cap from the pen prior to use. | n | xx |
| | Easily [1] | XX (XX%) |
| | With some difficulty [2] | XX (XX%) |
| | Did not complete [3] | XX (XX%) |
| Check that the subject / caregiver injects within 5 minutes of removing the needle cap. | n | XX |
| • | Easily [1] | XX (XX%) |
| | With some difficulty [2] | XX (XX%) |
| | Did not complete [3] | XX (XX%) |
| Check that the subject / caregiver positions the pen straight on the injection site with the yellow needle guard flat on the skin. | n | XX |
| | Easily [1] | XX (XX%) |
| | With some difficulty [2] | XX (XX%) |
| | Did not complete [3] | XX (XX%) |

<sup>[1]</sup> Subject / caregiver completed task easily without repeated reference to the IFU.

Note: If a subject has more than one attempt to self-administer study treatment at a single visit, only the first attempt is included in this summary.

<sup>[2]</sup> Subject / caregiver completed task but with some difficulty or repeated reference to the IFU for assistance.

<sup>[3]</sup> Subject / caregiver was not able to (or did not) complete task after multiple attempts and reference to the IFU, or intervention was required.

204959


Liquid Autoinjector

Example TAB\_INJ3 (cont.)

Protocol: 204959

Population: All Subjects (Safety)

# Table X.X Summary of Observer Checklist for In-Clinic Injections Autoinjector with Standard Label + Pictogram

Visit: WEEK 0

| | | (N=XX) |
|---|---|---|
| Check that the subject / caregiver starts the injection by pushing the pen all the way down. | n | XX |
| | Easily [1] | XX (XX%) |
| | With some difficulty [2] | XX (XX%) |
| | Did not complete [3] | XX (XX%) |
| Check that the subject / caregiver keeps the pen in position and pushes all the way down until a full dose is administered. | n | XX |
| | Easily [1] | XX (XX%) |
| | With some difficulty [2] | XX (XX%) |
| | Did not complete [3] | XX (XX%) |

- [1] Subject / caregiver completed task easily without repeated reference to the IFU.
- [2] Subject / caregiver completed task but with some difficulty or repeated reference to the IFU for assistance.
- [3] Subject / caregiver was not able to (or did not) complete task after multiple attempts and reference to the IFU, or intervention was required.

Note: If a subject has more than one attempt to self-administer study treatment at a single visit, only the first attempt is included in this summary.

userid: /arenv/arprod/compound/study/final/drivers/drivername.sas DDMMMYYYY HH:MM Programming Note: Continue for Week 8.


Timuid Autoinicator

Example TAB\_INJ4
Protocol: 204959

Population: All Subjects (Safety)

## 

Autoinjector with Standard Label + Pictogram

| | | Liquid Autoinjector<br>(N=XX) |
|---|---|---|
| User who logged in to complete the at-home injection checklist." | n | XX |
| | Patient | XX (XX%) |
| | Caregiver | XX (XX%) |
| Time from removal of pen from storage to injection (mins) | n | XX |
| | Mean | XX.X |
| | SD | XX.XX |
| | Median | XX.X |
| | Minimum | XX |
| | Maximum | XX |
| Did you need to contact the investigator / site prior to the injection for additional training? | n | XX |
| | Yes - Telephone | XX (XX%) |
| | Yes - Clinic Visit | XX (XX%) |
| | No | XX (XX%) |
| Was the pen stored in the fridge at 2-8 degrees C before preparing for use? | n | XX |
| 101 436. | Yes | XX (XX%) |
| | No | XX (XX%) |

<sup>[1]</sup> I was able to complete the task easily without repeated reference to the IFU.

<sup>[2]</sup> I was able to complete the task but with some difficulty or repeated reference to the IFU for assistance.

<sup>[3]</sup> I was not able to (or did not) complete task after multiple attempts and reference to the IFU.

Note: If a subject has more than one attempt to self-administer study treatment, only the first attempt is included in this summary.

204959

Example TAB\_INJ4 (cont.)

Protocol: 204959

Population: All Subjects (Safety)


# Table X.X Summary of Subject Completed Checklist for At-Home Injection at Week 4 Autoinjector with Standard Label + Pictogram

Liquid Autoinjector (N=XX)Check expiration date on the pen has not passed. XX n Easily [1] XX (XX%) With some difficulty [2] XX (XX%) Did not complete [3] XX (XX%) Look in the inspection window to check that the liquid is clear XX n (free from cloudiness or particles) and colorless to slightly yellow in color. Easily [1] XX (XX%) With some difficulty [2] XX (XX%) Did not complete [3] XX (XX%)

- [1] I was able to complete the task easily without repeated reference to the IFU.
- [2] I was able to complete the task but with some difficulty or repeated reference to the IFU for assistance.
- [3] I was not able to (or did not) complete task after multiple attempts and reference to the IFU.

Note: If a subject has more than one attempt to self-administer study treatment, only the first attempt is included in this summary.

204959

Example TAB\_INJ4 (cont.)

Protocol: 204959

Population: All Subjects (Safety)


## 

| | | Liquid Autoinjector<br>(N=XX) |
|---|---|---|
| Remove the clear needle cap from the pen by pulling it straight off. | n | XX |
| | Easily [1] | XX (XX%) |
| | With some difficulty [2] | XX (XX%) |
| | Did not complete [3] | XX (XX%) |
| Inject within 5 minutes of removing the needle cap. | n | XX |
| | Easily [1] | XX (XX%) |
| | With some difficulty [2] | XX (XX%) |
| | Did not complete [3] | XX (XX%) |
| Position the pen straight on the injection site with the yellow needle guard flat on the skin as show. | n | XX |
| | Easily [1] | XX (XX%) |
| | With some difficulty [2] | XX (XX%) |
| | Did not complete [3] | XX (XX%) |

<sup>[1]</sup> I was able to complete the task easily without repeated reference to the IFU.

Note: If a subject has more than one attempt to self-administer study treatment, only the first attempt is included in this summary.

<sup>[2]</sup> I was able to complete the task but with some difficulty or repeated reference to the IFU for assistance.

<sup>[3]</sup> I was not able to (or did not) complete task after multiple attempts and reference to the IFU.

204959

Example TAB\_INJ4 (cont.)

Protocol: 204959

Population: All Subjects (Safety)


# Table X.X Summary of Subject Completed Checklist for At-Home Injection at Week 4 Autoinjector with Standard Label + Pictogram

| | | Liquid Autoinjector (N=XX) |
|---|---|---|
| To start the injection, push the pen all the way down and hold. | n | XX |
| | Easily [1] | XX (XX%) |
| | With some difficulty [2] | XX (XX%) |
| | Did not complete [3] | XX (XX%) |
| Pen is kept in position and pushed all the way down until a full dose is administered. | n | XX |
| | Easily [1] | XX (XX%) |
| | With some difficulty [2] | XX (XX%) |
| | Did not complete [3] | XX (XX%) |

Note: If a subject has more than one attempt to self-administer study treatment, only the first attempt is included in this summary.

<sup>[1]</sup> I was able to complete the task easily without repeated reference to the IFU.

<sup>[2]</sup> I was able to complete the task but with some difficulty or repeated reference to the IFU for assistance.

<sup>[3]</sup> I was not able to (or did not) complete task after multiple attempts and reference to the IFU.

204959


Example TAB\_INJ5
Protocol: 204959

Population: All Subjects (Safety)

Table X.X
Summary of Device Usability/Functionality Questionnaire
Autoinjector with Standard Label + Pictogram

| Question | Category | Liquid Autoinjector (N=XX) |
|---|---|---|
| How comfortable did you feel with the training you received on how to use the autoinjector to administer your Nucala (mepolizumab)? | n | XX |
| | Not at all comfortable | XX (XX%) |
| | A little comfortable | XX (XX%) |
| | Moderately comfortable | XX (XX%) |
| | Very comfortable | XX (XX%) |
| | Extremely comfortable | XX (XX%) |
| At the end of the study, how confident were you about your ability to use the autoinjector in the correct way on your own when you were not in the doctor's office? | n | XX |
| | Not at all confident | XX (XX%) |
| | A little confident | XX (XX%) |
| | Moderately confident | XX (XX%) |
| | Very confident | XX (XX%) |
| | Extremely confident | XX (XX%) |

Programming Note: Continue for all remaining questions on the questionnaire.

Example TAB\_PD1 Protocol: 204959

Protocol: 204959 
Population: Pharmacodynamic

Table X

Summary of Blood Eosinophils (GI/L) by Visit

Treatment: Liquid Autoinjector (N=XX)

| Visit | n | Geom.<br>Mean | 95% CI<br>(Lower,Upper) | SD (logs) | Min. | Median | Max. |
|---|---|---|---|---|---|---|---|
| SCREENING | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xxx | XX.X | xxxx.xx | xx.x |
| WEEK 0 | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | xxxx.xx | XX.X |
| WEEK 4 | XX | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| WEEK 8 | XX | XXXX.XX | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| WEEK 12 | XX | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |

204959

Example TAB\_PD2 Protocol: 204959

Protocol: 204959 
Population: Pharmacodynamic

Table X

Summary of Ratio to Baseline Blood Eosinophils by Visit

Treatment: Liquid Autoinjector (N=XX)

| *** | | Geom. | 95% CI | an (1 ) | 261 | 26 11 | ., |
|---|---|---|---|---|---|---|---|
| Visit | n | Mean | (Lower, Upper) | SD (logs) | Min. | Median | Max. |
| WEEK 4 | XX | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| WEEK 8 | XX | XXXX.XX | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| WEEK 12 | XX | XXXX.XX | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |

Example TAB\_PD3 Protocol: 204959

Protocol: 204959 

Population: Pharmacodynamic

Table X

Summary of Blood Eosinophils (GI/L) by Visit and Baseline Mepolizumab Use

Treatment: Liquid Autoinjector (N=XX)

| Baseline Mepolizumab Use | N | Visit | n | Geom.<br>Mean | 95% CI<br>(Lower,Upper) | SD (logs) | Min. | Median | Max. |
|---|---|---|---|---|---|---|---|---|---|
| Yes | XX | SCREENING<br>WEEK 0<br>WEEK 4<br>WEEK 8<br>WEEK 12 | XX<br>XX<br>XX<br>XX<br>XX | xxxx.xx<br>xxxx.xx<br>xxxx.xx<br>xxxx.xx | (xxxx.xx,xxxx.xx)<br>(xxxx.xx,xxxx.xx)<br>(xxxx.xx,xxxx.xx)<br>(xxxx.xx,xxxx.xx)<br>(xxxx.xx,xxxx.xx) | xx.xxx<br>xx.xxx<br>xx.xxx<br>xx.xxx | XX.X<br>XX.X<br>XX.X<br>XX.X | xxxx.xx<br>xxxx.xx<br>xxxx.xx<br>xxxx.xx | xx.x<br>xx.x<br>xx.x<br>xx.x<br>xx.x |
| No | XX | SCREENING<br>WEEK 0<br>WEEK 4<br>WEEK 8<br>WEEK 12 | XX<br>XX<br>XX<br>XX<br>XX | xxxx.xx<br>xxxx.xx<br>xxxx.xx<br>xxxx.xx | (xxxx.xx,xxxx.xx)<br>(xxxx.xx,xxxx.xx)<br>(xxxx.xx,xxxx.xx)<br>(xxxx.xx,xxxx.xx)<br>(xxxx.xx,xxxx.xx) | xx.xxx<br>xx.xxx<br>xx.xxx<br>xx.xxx | XX.X<br>XX.X<br>XX.X<br>XX.X | xxx.xx<br>xxx.xx<br>xxx.xx<br>xxx.xx | xx.x<br>xx.x<br>xx.x<br>xx.x<br>xx.x |

204959

Example TAB\_PD4
Protocol: 204959

Protocol: 204959

Population: Pharmacodynamic

Table X

Summary of Ratio to Baseline Blood Eosinophils by Visit and Baseline Mepolizumab Use

Treatment: Liquid Autoinjector (N=XX)

| Baseline Mepolizumab Use | N | Visit | n | Geom.<br>Mean | 95% CI<br>(Lower,Upper) | SD (logs) | Min. | Median | Max. |
|---|---|---|---|---|---|---|---|---|---|
| Yes | XX | WEEK 4<br>WEEK 8<br>WEEK 12 | XX<br>XX<br>XX | xxxx.xx<br>xxxx.xx<br>xxxx.xx | (xxxx.xx,xxxx.xx)<br>(xxxx.xx,xxxx.xx)<br>(xxxx.xx,xxxx.xx) | xx.xxx<br>xx.xxx<br>xx.xxx | XX.X<br>XX.X<br>XX.X | XXXX.XX<br>XXXX.XX | xx.x<br>xx.x<br>xx.x |
| No | XX | WEEK 4<br>WEEK 8<br>WEEK 12 | XX<br>XX<br>XX | xxxx.xx<br>xxxx.xx<br>xxxx.xx | (xxxx.xx,xxxx.xx)<br>(xxxx.xx,xxxx.xx)<br>(xxxx.xx,xxxx.xx) | xx.xxx<br>xx.xxx<br>xx.xxx | xx.x<br>xx.x<br>xx.x | xxxx.xx<br>xxxx.xx | xx.x<br>xx.x<br>xx.x |

Example TAB\_S1
Protocol: 20495

Protocol: 204959 Page 1 of 3

Population: All Subjects (Safety)

#### Table X.X

Summary Profile of On-Treatment Adverse Events Defined by the Investigator as Allergic (Type I Hypersensitivity) Reactions

| | | Liquid Autoinjector (N=XX) |
|---|---|---|
| 1 | All Events | |
| | >= 1 event [1] | xx/xx (x%) |
| | 1 event | xx (x%) |
| | 2 events | xx (x%) |
| | 3 events | xx (x%) |
| | >=4 events | xx (x%) |
| 2 | <pre>Serious Events &gt;= 1 event [1]</pre> | xx/xx (x%) |
| 3 | Events considered related to investigational product >= 1 event [1] | xx/xx (x%) |
| 3.5 | Events reported on the day of dosing >= 1 event [1] | xx/xx (x%) |
| 4 | Intensity [1] | |
| | Mild | xx/xx (x%) |
| | Moderate | xx/xx (x%) |
| | Severe | xx/xx (x%) |
| 5 | Outcome [1] | |
| | Recovered/Resolving | xx/xx (x%) |
| | Recovering/Resolving | xx/xx (x%) |
| | Not recovered/Not Resolved | xx/xx (x%) |
| | Recovered/Resolved with sequelae | xx/xx (x%) |
| | Fatal | xx/xx (x%) |

<sup>[1]</sup> Information presented as number of events / number (%) subjects with at least one event. Subjects may be counted in more than one row.

<sup>[2]</sup> Cardiac History=Yes includes all subjects with any past medical condition under Cardiac Disorders.

<sup>[3]</sup> Unable to categorise time since last dose as event time not reported.

204959

Example TAB\_S1 (Cont.)

Protocol: 204959

Population: All Subjects (Safety)

#### Table X.X

Summary Profile of On-Treatment Adverse Events Defined by the Investigator as Allergic (Type I Hypersensitivity) Reactions

| | | Liquid Autoinjector<br>(N=XX) |
|----|--------------------------------|-------------------------------|
| 6 | Action Taken [1] | , , |
| | Study treatment withdrawn | xx/xx (x%) |
| | Dose reduced | xx/xx (x%) |
| | Dose increased | xx/xx (x%) |
| | Dose not changed | xx/xx (x%) |
| | Dose interrupted/delayed | xx/xx (x%) |
| | Not applicable | xx/xx (x%) |
| 7 | Cardiac History [1][2] | |
| | Yes | xx/xx (x%) |
| | No | xx/xx (x%) |
| 8 | Anaphylaxis Criteria Met | |
| | Anaphylactic Criterion 1 | xx/xx (x%) |
| | Anaphylactic Criterion 2 | xx/xx (x%) |
| | Anaphylactic Criterion 3 | xx/xx (x%) |
| 9 | No. doses prior to event [1] | |
| | 1 | xx/xx (x%) |
| | 2 | xx/xx (x%) |
| | 3 | xx/xx (x%) |
| | etc. | |
| 10 | No. doses prior to first event | |
| | 1 | xx (x%) |
| | 2 | xx (x%) |
| | 3 | xx (x%) |
| | etc. | |

<sup>[1]</sup> Information presented as number of events / number (%) subjects with at least one event. Subjects may be counted in more than one row.

<sup>[2]</sup> Cardiac History=Yes includes all subjects with any past medical condition under Cardiac Disorders.

 $<sup>\[3\]</sup>$  Unable to categorise time since last dose as event time not reported.

204959

Example TAB\_S1 (Cont.)

Protocol: 204959 Page 3 of 3

Population: All Subjects (Safety)

#### Table X.X

Summary Profile of On-Treatment Adverse Events Defined by the Investigator as Allergic (Type I Hypersensitivity) Reactions

| | | Liquid Autoinjector (N=XX) |
|----|-------------------------------------------|----------------------------|
| 11 | Time since last dose to event onset [1] | |
| | <=1 hr | xx/xx (x%) |
| | 1-<6 hrs | xx/xx (x%) |
| | 6-<24 hrs | xx/xx (x%) |
| | >=24 hrs | xx/xx (x%) |
| | Missing [3] | xx/xx (x%) |
| 12 | Time since last dose to first event onset | |
| | <=1 hr | xx (x%) |
| | 1-<6 hrs | xx (x%) |
| | 6-<24 hrs | xx (x%) |
| | >=24 hrs | xx (x%) |
| | Missing [3] | xx (x%) |
| 13 | No. symptoms associated with event [1] | |
| | 0 symptoms | xx/xx (x%) |
| | 1 symptom | xx/xx (x%) |
| | 2-5 symptoms | xx/xx (x%) |
| | >5 symptoms | xx/xx (x%) |
| 14 | Symptoms [1] | |
| | ABDOMINAL | xx/xx (x%) |
| | ANGIOEDEMA | xx/xx (x%) |
| | ARTHRALGIA<br>Etc. | xx/xx (x%) |
| | ELC. | |

- [1] Information presented as number of events / number (%) subjects with at least one event. Subjects may be counted in more than one row.
- [2] Cardiac History=Yes includes all subjects with any past medical condition under Cardiac Disorders.
- [3] Unable to categorise time since last dose as event time not reported.

204959

#### Programming Notes: -

Remove footnotes that are not relevant for the table.

Sections 1 - 6, 9, 10: Create for all adverse events of special interest

Sections 9 and 10: For studies longer than 1 year can consider the following categories: 1, 2, 3, 4, 5, 6, 7-12, 13-18,

19-24, >24

Section 7: Only for the following adverse events of special interest

Serious Cardiac, Vascular and Thromboembolic Events

Serious Ischemic Events

Section 8: Only for the following adverse events of special interest

Anaphylaxis

Systemic - Allergic (Type I Hypersensitivity)

Sections 11 - 14: Only for the following adverse events of special interest

Anaphylaxis

Systemic - Allergic (Type I Hypersensitivity) and Other Systemic

Systemic - Allergic (Type I Hypersensitivity)

Systemic - Other Systemic Local Injection Site Reactions

Section 3.5: Only for the following adverse events of special interest

Anaphylaxis

Systemic - Allergic (Type I Hypersensitivity) and Other Systemic

Systemic - Allergic (Type I Hypersensitivity)

Systemic - Other Systemic

Page 2 of 2

Example TAB\_S2
Protocol: 204959

Population: All Subjects (Safety)

Table X
Summary of Binding Antibody Results by Visit

| Visit | Assay Result | | Liquid Autoinjector (N=XX) |
|---|---|---|---|
| WEEK 0 | n | | X |
| HEER O | NEGATIVE | | X (XX%) |
| | POSITIVE | | X (XX%) |
| WEEK 12/EARLY WITHDRAWAL | n | | X |
| WEEK 12/EAKUI WIIIDKAWAL | NEGATIVE | | X (XX%) |
| | POSITIVE | | X (XX%) |
| | Titre value | Min.<br>Median<br>Max. | X<br>X.X<br>X |

204959

Example TAB\_S3
Protocol: 204959

Protocol: 204959 Page 1 of X

Population: All Subjects (Safety)

Table X

Summary of Injection Pain - VAS Scores (mm)

Treatment: Liquid Autoinjector (N=XX)

| Visit | N | Planned Relative Time | n | Mean | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|
| WEEK 0 | XX | INJECTION | XX | X.X | X.XX | X.X | XX | XX |
| | | 1 HR POST INJECTION | XX | X.X | X.XX | X.X | XX | XX |
| | | 24 HRS POST INJECTION | XX | X.X | X.XX | X.X | XX | XX |
| WEEK 4 | XX | INJECTION | XX | X.X | X.XX | X.X | XX | XX |
| | | 1 HR POST INJECTION | XX | X.X | X.XX | X.X | XX | XX |
| | | 24 HRS POST INJECTION | XX | X.X | X.XX | X.X | XX | XX |
| WEEK 8 | XX | INJECTION | XX | X.X | X.XX | X.X | XX | XX |
| | | 1 HR POST INJECTION | XX | X.X | X.XX | X.X | XX | XX |
| | | 24 HRS POST INJECTION | XX | X.X | X.XX | X.X | XX | XX |

204959


Example TAB\_S4
Protocol: 204959

Population: All Subjects (Safety)

Table X

Summary of Injection Pain - Categorical Pain Assessment

Visit: WEEK 0 (N=XX)

| Planned<br>Relative Time | Pain Assessment | Category | Liquid Autoinjector<br>(N=XX) |
|---|---|---|---|
| INJECTION | VAS Score (mm) | n | XX |
| | | 0 | XX (XX%) |
| | | >0 | XX (XX%) |
| | Description of Pain [1] | n | XX |
| | | Sharp/Stinging | XX (XX%) |
| | | Dull/aching | XX (XX%) |
| | | Burning | XX (XX%) |
| | | Other | XX (XX%) |
| | Pain Relative to Expectation | n | XX |
| | | Greater than expected | XX (XX%) |
| | | Less than expected | XX (XX%) |
| | | As expected | XX (XX%) |
| | Pain acceptable? | n | XX |
| | - | Yes | XX (XX%) |
| | | No | XX (XX%) |

<sup>[1]</sup> More than one description may be ticked.

userid: /arenv/arprod/compound/study/final/drivers/drivername.sas DDMMMYYYY HH:MM

Programming Note: continue for planned relative time = 1 HR POST INJECTION, 24 HRS POST INJECTION and Week 4 and 8.

204959

Example TAB\_EX1
Protocol: 204959

Population: All Subjects Enrolled


Table X

Summary of Number of Subjects With at Least One On-Treatment Exacerbation

Liquid Autoinjector (N=XX)

Population

Number of Subjects With at Least One Exacerbation

XX (XX%)


Example TAB\_ECG1 Protocol: 204959

Population: All Subjects (Safety)

| | Population | Liquid Autoinjector<br>(N=XX) |
|------------------------------|--------------|-------------------------------|
| Baseline | _ | XX |
| bdseline | n a s | |
| | <=450 | XX (XX%) |
| | >450 - <=480 | XX (XX%) |
| | >480 - <=500 | XX (XX%) |
| | >500 | XX (XX%) |
| Week 12 | n | XX |
| | <=450 | XX (XX%) |
| | >450 - <=480 | XX (XX%) |
| | >480 - <=500 | XX (XX%) |
| | >500 | XX (XX%) |
| Week 12 Change from Baseline | N | XX |
| | <-60 | XX (XX%) |
| | >=-60 - <-30 | XX (XX%) |
| | >=-30 - <0 | XX (XX%) |
| | >=0 - <30 | XX (XX%) |
| | >=30 - <60 | XX (XX%) |
| | >=60 | XX (XX%) |

204959

Example LIST\_POP1

Protocol: 204959


Population: All Subjects (Safety)

Table X.X

Listing of Baseline Mepolizumab Use

Treatment: Liquid Autoinjector

Site Id./

| Unique<br>Subject Id. | | <u> </u> | Most Recent Blood Eosinophil Count Prior to Starting Mepolizumab (cells/uL)[2] |
|---|---|---|---|
| XXXXXX/<br>MID204959 XXXXXX | Yes | Yes | 300 |

<sup>[1]</sup> Blood eosinophil count immediately before starting mepolizumab that was >= 150 cells/uL or a blood eosinophil count that was >= 300 cells/uL in the 12 months prior to starting mepolizumab.

<sup>[2]</sup> Historical value taken prior to starting mepolizumab for subjects currently receiving treatment with mepolizumab only.

204959

Example LIST\_POP2 Protocol: 204959

Protocol: 204959 

Population: All Subjects (Safety)

Table X.X

Listing of Previous Mepolizumab Clinical Trials

Treatment: Liquid Autoinjector

| Site Id./<br>Unique<br>Subject Id. | Did the subject participate in a previous mepolizumab clinical trial? | Previous Protocol<br>Identifier | Previous Subject Number |
|---|---|---|---|
| XXXXXX/<br>MID204959.XXXXXX | Yes | 205667 | XXX |

204959

Example LIST\_INJ1 Protocol: 204959

Protocol: 204959 
Population: All Subjects (Safety)

Was Self-

Table X.X

Listing of Investigator Assessment of Injection Success

Treatment: Liquid Autoinjector, Standard Label + Pictogram

Visit/

| Site Id./<br>Unique<br>Subject Id. | | Date of<br>Assessment | Administration of Injection Successful? | User Error | Device Error |
|---|---|---|---|---|---|
| XXXXXX/<br>MID204959.XXXXXX | WEEK 0/<br>IN-CLINIC | DDMMYYYY | Yes | | |
| | WEEK 4/<br>HOME | DDMMYYYY | Yes | | |
| | WEEK 8/<br>IN-CLINIC | DDMMYYYY | Yes | | |
| XXXXXX/<br>MID204959.XXXXXX | WEEK 0/<br>IN-CLINIC | DDMMYYYY | No | Incorrect injection site selected - arm | |
| | UNSCHED/<br>IN-CLINIC | DDMMYYYY | Yes | | |
| XXXXXX/<br>MID204959.XXXXXX | WEEK 0/<br>IN-CLINIC | DDMMYYYY | No | | Syringe leaking<br>Components broken / cracked |

Example LIST\_INJ2

Protocol: 204959 

Population: All Subjects (Safety)

Table X.X

Listing of Person Administering Injection [1] and Time From Removal of Syringe from Storage to Injection

Treatment: Liquid Autoinjector

| Site Id./<br>Unique<br>Subject Id. | Visit | Confirm who will be administering the injection [1] | Time from removal of autoinjector from storage to injection (mins) |
|---|---|---|---|
| XXXXXX/<br>MID204959.XXXXXX | WEEK 0 | Patient | Yes |
| 1112201303,11111111111 | WEEK 4 | Patient | Yes |
| | WEEK 8 | Patient | Yes |
| XXXXXX/<br>MID204959.XXXXXX | WEEK 0 | Patient | Yes |

<sup>[1]</sup> For the at-home injection (week 4), the person administering the injection is documented by the eDiary as the user (caregiver/patient) who logged in to complete the at-home injection checklist.

Note: If a subject has more than on attempt to self-administer study treatment, only information for the first attempt is available in the eDiary.

204959

Example LIST\_EX1 Protocol: 204959

Protocol: 204959 

Population: All Subjects (Safety)

Table X.X Listing of Exacerbations

Treatment: Liquid Autoinjector

| Site<br>Id. | Unique Subject Id. | Date of<br>Onset | Treatment<br>Phase | Withdrawn | Outcome/<br>End Date | CS<br>Taken [1] | Hospitalised?/<br>ER Visit? | Intubated? |
|---|---|---|---|---|---|---|---|---|
| PPD | MID204959.XXXXXX | DDMMYYYY | On-Treatment | No | RESOLVED/<br>DDMMYYYY | Y | N/<br>N | N |

userid: /arenv/arprod/compound/study/final/drivers/drivername.sas DDMMMYYYY HH:MM

[1] CS = Systemic/oral corticosteroids

204959

Example LIST\_S1 Protocol: 204959

Protocol:  $20\overline{4}959$  

Population: All Subjects (Safety)

Table X.X Listing of Injection Pain Assessment

Treatment: Liquid Autoinjector

| Site Id./ | Visit/ | | | VAS | | | Was the |
|---|---|---|---|---|---|---|---|
| Unique | Planned | Date/Time of | Study | Score | | Pain Relative | Pain |
| Subject Id. | Relative Time | Assessment | Day | (mm) | Description of pain | to Expectation | Acceptable? |
| XXXXXX/<br>MID204959.XXXXXX | WEEK 0/<br>INJECTION | DDMMYYYY/<br>HH:MM | 1 | XX | Sharp/stinging | Greater | Yes |

204959

Example LIST\_PD1 Protocol: 204959

Protocol: 204959

Population: Pharmacodynamic

Table X.X

Listing of Blood Eosinophils (units)

Treatment: Liquid Autoinjector

| Site Id./<br>Unique<br>Subject Id. | Age (years)/<br>Sex/<br>Race | Visit | Date/<br>Study Day | Result | Change from<br>Baseline | Ratio to<br>Baseline | Normal Range | NR Flag |
|---|---|---|---|---|---|---|---|---|
| XXXXXX/<br>MID204959.XXXXXX | XX/<br>F/<br>ASIAN | WEEK 0 | YYYY-MM-DD/<br>1 | XX.XX | XX.XX | X.XX | x.xx - x.xx | NORMAL |

<sup>[1]</sup> NR = Normal Range.

Example FIG\_PD1

Protocol: 204959

Population: Pharmacodynamic

Figure X.X Geometric Mean Ratio to Baseline Blood Eosinophils by Visit and Baseline Mepolizumab Use

